# The ENRGISE Pilot Study Protocol

## 1. Project Title:

The ENRGISE Pilot Study

# 2. Investigators

Dual PI grant: Marco Pahor PI (ACC)

Walter Ambrosius PI (DMAQC)

DMAQC: Michael Miller, Mark Espeland, Daniel Beavers, Kristina Lewis

Biorepository: Russell Tracy

ACC: Christiaan Leeuwenburgh, Samuel Wu

Field Centers

Wake Forest School of Medicine: Stephen Kritchevsky

University of Florida: Todd Manini, Stephen Anton

Northwestern University: Mary McDermott

Tufts University: Roger Fielding, Christine Liu University of Pittsburgh: Anne Newman, Jane Cauley

# 3. Abstract

Growing evidence shows that low-grade chronic inflammation, characterized by elevations in plasma C-reactive protein, tumor necrosis factor alpha, and particularly Interleukin-6 (IL-6), is an independent risk factor of disability, impaired mobility, and lower walking speed. Low-grade chronic inflammation is a modifiable risk factor. However, it is unknown whether interventions that reduce the levels of inflammatory markers *per se* improve mobility, or avert decline in mobility in older persons.

To address this gap in evidence we conduct the randomized clinical trial ENRGISE (ENabling Reduction of low-Grade Inflammation in SEniors) Pilot Study to test the ability of anti-inflammatory interventions for preventing major mobility disability by improving or preserving walking ability. We have maximized the public health impact by selecting interventions that are safe, tolerable, acceptable, and affordable for vulnerable older persons. Specifically, in this trial we test the efficacy vs. placebo of the angiotensin receptor blocker losartan and omega-3 polyunsaturated fatty acids in the form of fish oil, alone and in combination. Both angiotensin receptor blockers and omega-3 polyunsaturated fatty acids have shown to reduce IL-6 in clinical trials and preliminary data suggest that they may improve physical function.

We recruit older persons who are at risk for, or with, mobility impairment, as measured by slow gait speed and self-reported mobility difficulty, and who have elevated levels of IL-6, the marker most consistently associated with mobility limitations. Preliminary data regarding feasibility need to be gathered before such a trial can be effectively designed and implemented. We conduct The ENRGISE Pilot Study to assess the effects of the interventions on several inflammatory markers, walking speed, physical function and strength. This allows us to refine the design, recruitment yields, target population, adherence, retention, tolerability, sample-size, and cost for the main ENRGISE trial.

# 4. Specific aims

Growing evidence from our group and others shows that low-grade chronic inflammation, characterized by elevations in plasma C-reactive protein (CRP), tumor necrosis factor Alpha (TNF- $\alpha$ ), and particularly interleukin-6 (IL-6), 1-7 is an independent risk factor for disability, impaired mobility, and slow walking speed. Low-grade chronic inflammation is a modifiable risk factor. However, it is unknown whether interventions that reduce the levels of inflammatory markers *per* se improve mobility, or avert decline in mobility in older persons.

To address this gap in evidence, we will conduct the main randomized clinical trial (RCT) **ENRGISE** (**ENabling Reduction of low-Grade Inflammation in SEniors**) to test the ability of anti-inflammatory interventions for improving or preserving walking ability. We have maximized the <u>public health impact</u> of the interventions by selecting interventions that are safe, tolerable, acceptable, and affordable for vulnerable older persons. Based on an extensive literature review, we test the efficacy of the angiotensin receptor blocker (ARB) losartan (LO) and omega-3 polyunsaturated fatty acids (ω-3) as fish oil. To maximize the anti-inflammatory effect and potential benefit on mobility, we explore both individual and combination interventions that target different, but complementary and potentially synergistic anti-inflammatory mechanisms. <sup>12-15</sup> We plan to recruit older persons at risk for, or with, mobility impairment, as measured by <u>slow gait speed and self-reported mobility difficulty</u>, and who have elevated blood levels of <u>IL-6 (>2.5 pg/ml)</u>, the marker most consistently associated with mobility limitations. <sup>1-7</sup> Preliminary data on feasibility and information required for obtaining sample size estimates are needed to effectively design and implement the main trial. Thus, we implement the following **specific aims** for the ENRGISE Pilot Study:

- a. Conduct a pilot RCT in 300 older persons at risk of mobility decline to assess: (i) compared with placebo, the effects of LO,  $\omega$ -3, and LO+ $\omega$ -3 on IL-6 and walking speed; (ii) the recruitment yields, the target population, adherence, retention, tolerability, sample-size, design, and cost for the main RCT; and (iii) the intra-subject variability of IL-6, and the dosage and safety of the interventions.
- b. Measure novel and established inflammatory markers to:
  - i. Characterize the effect of LO and  $\omega$ -3 on these biomarkers and determine: (a) Are these cytokines/pathways impacted by the interventions? (b) Are the changes in these markers pre- vs. post-intervention less than, equivalent to, or greater than that of IL-6? and
  - ii. Assess if these biomarkers yield independent information from IL-6 with respect to change in walking speed and/or provide benefit for screening participants for the main trial.

ENRGISE addresses critical public health issues regarding mobility disability prevention. We test the antiinflammatory effects of widely available inexpensive interventions and their impact on mobility in a highly vulnerable population of older adults at risk of mobility disability.

#### 5. Background

**Mobility outcomes.** Preserving mobility is central to maintaining a high quality of life and participation in activities to be fully independent in the community. <sup>16, 17</sup> Mobility limitation is associated with subsequent hospitalization, nursing home placement, increased healthcare costs, and death. <sup>18-22</sup>

**Low-grade chronic inflammation and mobility outcomes.** Acute inflammation is tightly regulated to promote healing and response to infection. In young, healthy persons, levels of inflammatory markers are low, while many older adults, even if apparently disease-free, have persistent, chronic, mild elevations of CRP, IL-6, TNF- $\alpha$ , and other markers. The degree of these elevations predicts disability, mobility limitations<sup>1, 3</sup> and mortality<sup>23-25</sup> independently of other risk factors. The basis for these elevations in older adults is not well understood. Smoking history and obesity,<sup>26</sup> especially visceral adiposity,<sup>26</sup> play a role, yet age itself remains the strongest predictor of these elevations in inflammatory markers.<sup>1</sup> Studies of the aging process suggest that senescent cells secrete IL-6, initiated by IL-1 $\alpha$  and regulated by TGF $\beta$ .<sup>27</sup> Due to cell cycle arrest, senescent cells are less prone to malignant transformation, but may disrupt normal tissue function, promoting central adiposity, atherosclerotic plaque, and osteoporosis.<sup>27, 28</sup> Reduced renal function<sup>29</sup> and atherosclerosis<sup>30, 31</sup> may contribute

to the elevation of inflammatory markers, through decreased excretion and increased production of these markers. Thus, the "chronic inflammation" of aging may indicate the ongoing process of age-related damage and repair, and thus, contribute to the cumulative burden of disease-related damage, and cellular senescence.

The age-related dysregulation of immune function may have direct adverse consequences on physical function and promote disability by causing fatigue and loss of muscle strength. <sup>7, 32, 33</sup> CRP has been identified as an independent risk factor for cardiovascular disease (CVD) outcomes, <sup>34-38</sup> and clinical trials targeting the up-regulation of inflammation to reduce CVD events are currently underway. <sup>39-41</sup> In aging, IL-6 is thought to have a direct impact on fatigue and loss of muscle function. Injection of IL-6 produces acute and chronic atrophy of skeletal muscle in rats. <sup>42</sup> IL-6 levels tracked best with functional decline, <sup>1, 4</sup> though many inflammatory markers are involved and related to frailty. <sup>43, 44</sup> While conditions, such as myocardial infarction, stroke and arthritis, may contribute to disability and inflammation, the inflammatory state appears to have a direct downstream causal effect on disability. It follows that treatments that moderate the inflammatory pathway and reduce IL-6 may ameliorate mobility. Inflammatory pathways are tightly regulated so that manipulation could have adverse effects such as infection or delay of healing. Though exercise and weight loss both reduce IL-6 levels and improve mobility function providing circumstantial support, <sup>45, 46</sup> to our knowledge, the hypothesis that IL-6 reduction improves mobility function has not been directly tested.

**Figure 5.1.** The relation of inflammation to loss of physical function. The three main sources of inflammation in the elderly (genetic and epigenetic factors, exogenous factors and endogenous factors) combine to cause molecular and biochemical changes with important consequences, which in turn lead to physiological consequences, and ultimately to mobility limitation and mortality. These changes are complex with thousands of genes and other macromolecules involved; some examples of important pathways are listed. The potential impact of the chosen interventions are shown.



**Detrimental mechanisms of action of inflammation in older persons.** The sources and consequences of chronic inflammation are important for identifying promising interventions (Figure 5.1.). Inflammation in older persons results from: genes and their modifiers, the environment, and the *in situ* biochemical environment. Important exogenous environments include smoking, moderate (beneficial) and excessive alcohol consumption, and an anti-oxidative diet (beneficial). Pro-inflammatory endogenous factors include adiposity (especially visceral adiposity), subclinical disease burden, and oxidative stress, among others.

Regarding direct consequences, activation of NF- $\kappa$ B signaling increases muscle protein degradation and inhibits myogenesis, 47, 48 except in very late differentiation where it promotes homeostasis. 47 NLRP3-mediated IL-1 $\beta$  production plays a major role in mediating age-associated inflammation; ablation of this complex improves inflammation-associated detrimental changes with aging. 49 This inflammosome is activated by several products of damage including certain free fatty acids, free cholesterol, and reactive oxygen species. 49

The cytokines TNF- $\alpha$  and IL-1 $\beta$  inhibit hormones critical for muscle homeostasis (e.g., growth hormone and IGF-1).<sup>47</sup> Circulating IL-6 is negatively associated with myosin heavy chain synthesis in patients with heart failure.<sup>50</sup> TNF- $\alpha$  activates muscle matrix metalloproteinase-9 (MMP-9), which degrades the extracellular matrix,<sup>51</sup> and can cause muscle cell apoptosis, which is attenuated by caloric restriction.<sup>52</sup> Cytokines also augment muscle infiltration by proinflammatory macrophage and lymphocytes,<sup>47</sup> including proinflammatory senescence-associated secretory phenotype (SASP) cells.<sup>53</sup> Aging muscle has accelerated mitochondriamediated apoptosis and mitophagy linked to increased oxidative stress.<sup>54</sup>

 $\omega$ -3 fatty acids are indicated to reduce triglyceride levels in adults with severe hypertriglyceridemia.  $\omega$ -3 fatty acids are also anti-inflammatory <sup>55</sup> via a specific  $\omega$ -3 fatty acid receptor, GP120 <sup>56</sup> which blocks NF- $\kappa$ B and JNK signaling, counter to saturated fatty acid-mediated proinflammatory TLR2 signaling. <sup>57</sup> Saturated fats

are generally pro-inflammatory,  $^{58}$  and can cause a decline in muscle protein synthesis via ER stress.  $^{59}$   $\omega$ -3 supplementation down-regulates inflammation in part through decreased TNF- $\alpha$  expression and  $\omega$ -3 fatty acids are likely to improve mTOR signaling, thereby stimulating muscle protein synthesis in humans.  $^{61}$  A meta-analysis of several RCTs has shown that  $\omega$ -3 reduce both IL-6 and CRP in chronic non-autoimmune disease.  $^{62}$ 

ARBs are primarily indicated for the treatment of hypertension. The ARB LO is also a partial PPAR- $\gamma$  agonist,  $^{63}$  yielding potent anti-inflammatory effects.  $^{64}$  LO reduces IL-6 in human  $^{65}$  and animal studies,  $^{66}$  possibly through PPAR- $\gamma$ /AMPK agonism, blockage of proinflammatory angiotensin II AT1 signaling, or both.  $^{64}$ ,  $^{67}$  ARBs mitigate lipopolysaccharide -mediated inflammation, and inhibit TNF- $\alpha$ -mediated endothelial Receptor for Advanced Glycosylation Endproduct (RAGE) expression.  $^{68}$  LO has been shown to improve skeletal muscle related activity measures in older mice.  $^{66}$ ,  $^{69}$  In summary, inflammation plays a major role in the loss of physical function through a wide variety of mechanisms, many of which offer interventional targets.

All drugs have multiple effects.  $LO^{63, 67, 70}$  and  $\omega$ -3, $^{71, 72}$  in addition to averting inflammation, also affect vasculature, coagulation, metabolism, and skeletal muscle, all of which may benefit mobility (Figure 5.1.). Testing these two different interventions that avert inflammation may provide added support regarding the relevance of their common anti-inflammatory effect in possibly benefiting walking speed and ultimately mobility. **Selection of anti-inflammatory interventions.** A broad range of pharmacological, nutritional, and behavioral

interventions have potential efficacy in reducing low grade chronic inflammation.<sup>39, 74</sup> To maximize the public health impact of ENRGISE, we set the criteria outlined in Table 5.1. and 5.2. for prioritizing interventions. Based on the selection criteria and the evidence reviewed below, in the pilot phase we test **LO and \omega-3**. Both have excellent safety records, are tolerable and acceptable, reduce elevated IL-6, have shown benefits in improving physical performance, have not been tested in similar trials, act with different but complementary biological mechanisms, 12-15 do not negatively interfere with neuromuscular metabolism, and are broadly available at low cost.  $\omega$ -3 reduced IL-6 by

Table 5.1. Criteria for prioritizing the selection of the ENRGISE interventions

- 1. <u>Safety, tolerability and acceptability</u> are key criteria. Vulnerable older persons use multiple drugs and have multiple comorbidities, and thus, are at high risk of adverse drug reactions. Newer drugs are often tested in younger or middle age adults for the treatment of a single condition and therefore, their safety and tolerability in older persons is not fully known.<sup>73</sup> Furthermore, for the prevention of mobility limitations, vulnerable or frail older persons may not be willing to take, and their providers may not be willing to prescribe drugs that bear a risk of severe adverse events. Finally, we exclude interventions that may <u>negatively affect</u> skeletal muscle or neuromuscular metabolism.
- 2. Reduction of IL-6 and possibly CRP in clinical trials is our primary criterion.
- Benefit on physical performance and/or skeletal muscle is a relevant, but not necessary criterion.
- 4. <u>Innovation</u>. We have prioritized interventions that have not been, or are not being tested in RCTs for preventing mobility limitations.
- 5. <u>Biological mechanisms</u> are considered to prioritize interventions that target different inflammatory mechanisms or may have synergistic effects. We exclude interventions that may negatively affect skeletal muscle metabolism.
- 6. <u>Practical and affordable</u> for implementation in the US health care system. <u>Cost</u> is a major factor for this criterion to maximize the public health impact of the trial

>50% in RCTs<sup>75, 76</sup> and ARBs reduced IL-6 by >40%<sup>77, 78</sup> and by 58%<sup>79</sup> in RCTs. In Health ABC¹ and EPESE,² we have found that a 50% lower IL-6 plasma level was associated with approximately 50% lower risk of mobility disability over 2.5 and 4 years of follow-up, respectively. Change in IL-6 induced by LO and  $\omega$ -3 may depend on the target population, baseline IL-6 level, dosage, compliance, and duration of treatment. Thus, the pilot study is of key importance to probe their anti-inflammatory effects in the ENRGISE population.

#### Inclusion of potential candidate interventions (see Table 5.2.)

Angiotensin Converting Enzyme Inhibitors (ACEIs) and ARBs have shown excellent safety in large hypertension and heart failure trials in older persons, <sup>80-84</sup> Among ACEIs, perindopril<sup>85, 86</sup> and enalapril<sup>65</sup> have demonstrated reductions in IL-6. Perindopril has shown to prevent physical function and walking speed decline in older persons, <sup>87</sup> to reduce CRP, <sup>88</sup> and to have a favorable safety profile. <sup>89</sup> Dual angiotensin blockade with ACEIs and ARB results in higher risk of adverse events, <sup>90</sup> thus, we do not recommend to combine ACEIs and ARBs. Virtually all ARBs, except azilsartan, have been shown to reduce elevated IL-6. <sup>65, 77, 91-102</sup> Telmisartan improved walking distance in patients with peripheral artery disease <sup>103</sup> and running endurance in mice. <sup>15</sup> In older mice LO reduced IL-6 and improved physical performance. <sup>66</sup> We prioritize ARBs because of greater tolerability than ACEIs, <sup>83, 84, 104</sup> and among ARBs, we prioritize LO due to its low cost (1/50 that of other ARBs). Among nutritionals, ω-3<sup>62</sup> and lipoic acid<sup>92, 105</sup> reduce IL-6<sup>62, 92, 105</sup> and CRP<sup>62, 106</sup> in RCTs. The evidence of the

anti-inflammatory effect is particularly strong for  $\omega$ -3. $^{62}$  In older women,  $\omega$ -3 improved walking speed, $^{107}$  and strength when supplemented to exercise. $^{108}$   $\omega$ -3 are widely available at low cost primarily in the form of fish oil. Among behavioral interventions, compared with Western diet, the Mediterranean diet (MED) reduces IL-6 $^{109\text{-}113}$  and CRP. $^{109,\,110,\,112,\,113}$  Olive oil contains oleocanthal acting as a natural anti-inflammatory compound that has a potency and profile similar to that of ibuprofen. $^{55,\,114}$  MED is associated with better physical performance, higher walking speed and lower risk of frailty. $^{115\text{-}118}$  MED is promising, however, after consulting with diet experts, including Dr. Linda Van Horn at NWU, Dr. Mara Vitolins at WFSM, and Dr. Stephen Anton at UF, it was concluded that diet interventions are complex and too resource intensive to be considered in this context, primarily due to the need for dietary counseling. Additionally, the most successful MED trials were conducted in Spain and Italy, $^{110,\,113,\,119}$  where MED is part of the local traditions. It is doubtful whether MED could be successfully imported in the ENRGISE older frail US population within the available resources of this trial. Thus, after careful consideration, we did not prioritize diet interventions.

#### **Exclusion of potential candidate interventions (see Table 5.2.)**

<u>Criterion #1</u> excludes anti-TNF- $\alpha$  agents (etanercept, infliximab, adalimumab), <sup>120</sup> anti-IL-6 agents (siltuximab), <sup>121</sup> anti-IL1 $\beta$  (canakinumab – no long-term safety data available), <sup>122</sup> and thiazolidinediones (rosiglitazone, pioglitazone) <sup>123</sup> for risk of infections, liver toxicity, fluid overload, CVD, fractures, or possible cancer. Chloroquine and statins are excluded due to concerns of myotoxicity <sup>124-126</sup> and lack of effect on walking speed for statins (Criteria #1, #5). <sup>127</sup> Corticosteroids, aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), and cyclooxygenase-2 (Cox-2) inhibitors are excluded for risk of bleeding, <sup>128-132</sup> gastrointestinal toxicity, and CV events for NSAIDs and COX-2 inhibitors. <sup>133</sup> Colchicine is excluded for risk of myotoxicity <sup>134, 135</sup> and neuropathy (Criteria #1, #5). <sup>135</sup> Low-dose methotrexate is potentially safe and effective in lowering IL-6. But, we found it is not acceptable by the older target population. A pilot study to assess effects on walking speed did not randomize a single participant, primarily because of refusal to take methotrexate expressed by participants or their health providers (section 3.d.3). Methotrexate bears the stigma of a "dangerous" anticancer drug in these older people. Many of the above excluded drugs would likely face similar non-acceptability problems; even if they were effective, they would have <u>limited public health impact for prevention</u>, due to high cost and risk of adverse effects.

<u>Criterion #2</u> excludes promising interventions, such as metformin, ghrelin, lactoferrin, oxytocin, salsalate, creatine, curcuma, probiotics, and resveratrol because of lack of clinical trial evidence of reducing IL-6. Metformin, while potentially promising, has shown in the DPP a small reduction in CRP (-12%), 136 in part related to its modest weight-reducing effect, however other trials have shown no effect on IL-6137 or CRP. 138-142

<u>Criterion #4.</u> Physical activity and weight loss have shown in multiple RCTs both reduction of IL-6 and prevention of mobility limitations, <sup>45, 46, 143-147</sup> and thus, are not prioritized as innovative approaches.

**Innovation and strengths.** The following features of ENRGISE represent innovative approaches:

- Targeting chronic low grade inflammation to achieve reduced inflammation and reduced mobility limitations
- Targeting an older population at high risk of mobility disability, which is often excluded from large RCTs
- Repurposing widely available inexpensive interventions (LO and ω-3)
- Table 5.2. Summary of selection criteria and candidate interventions (see details in the text) Criteria 1. Safe, 2. IL-6 3. Physical 4. Mecha Practical, tolerable. perforredu-Inno-Interventions acceptable affordable ction mance vation -nism ACEIs, ARBs + ນ-3 + Mediterranean diet + + + + + Physical activity, weight loss + + + \_ + +? Vitamin D + + + + + Anti-TNF- $\alpha$ , -IL6,-IL1; ? ? + methotrexate thiazolidinediones Statins, chloroquine, colchicine + - ? + + \_ \_ Corticosteroids, aspirin, + ? + + + \_ NSAIDs, cox-2 inhibitors Metformin, fosinopril, ghrelin, lactoferrin, oxytocin, salsalate, - ? - ? +? + curcuma, creatine, probiotics, resveratrol + positive evidence, - negative evidence, ? evidence lacking
- Testing LO and ω-3 in combination to maximize their effects on inflammation and mobility
- The use of several adaptive features in design and stratified screening for ENRGISE pilot study

The assessment of novel inflammatory markers in ENRGISE pilot study

#### 6. Research Plan

**6.1. Design.** We test LO,  $\omega$ -3 and their combination in a double-blind, placebo-controlled RCT (The ENRGISE Pilot Study). Randomization is concealed via the secure web-based data management system. We use a permuted block algorithm (with random block lengths).

LO and ω-3 are considered safe in elders. 80-84, 148, 149 We conduct this pilot RCT to (a) decide whether we should proceed to the main ENRIGISE trial with 1 or 2 interventions, and (b) if two interventions are warranted whether we should proceed as a three-arm (without the combination group) or a 2x2 factorial study. The pilot is designed to achieve the following goals: (1) estimate recruitment yields including percent consenting; (2) confirm safety and tolerability; (3) assess the impact of interventions on IL-6 and walking speed as well as the secondary outcomes of Short Physical Performance Battery (SPPB), frailty, and muscle strength; (4) evaluate the strength of relationship between the change in IL-6 with the change in walking speed; (5) allow selection of the interventions that demonstrate high participant compliance and retention; (6) collect data on outcomes of major mobility disability and other mobility measures; (7) support the decision to proceed with a factorial or parallel design; (8) examine intra-subject variability of IL-6; (9) explore the impact of the

interventions on additional biomarkers, their relationship with walking speed and their impact on recruitment and effect size estimates; and (10) estimate the cost of the main trial.

| Strata according to | LIFE | ENRGISE pilot | Randomization weights | | | |
|---|---|---|---|---|---|---|
| medication use at baseline | N (%) | N (%) | Placebo LO | LO | Placebo LO | LO |
| | Observed | Proposed | Placebo ω-3 | Placebo ω-3 | ω-3 | $\omega$ –3 |
| 1 No ω-3 (ACEI/ARB ok) | 637 (44.1) | 75 (25%) | 0.4* | 0 | 0.6* | 0 |
| 2 No ACEI/ARB (ω-3 ok) | 154 (10.7) | 75 (25%) | 0.4** | 0.6** | 0 | 0 |
| 3 No ACEI/ARB, No ω-3 | 655 (45.3) | 150 (50%) | 0.2 | 0.2 | 0.2 | 0.4 |
| Overall | | 300 (100%) | 0.3 (n=90) | 0.25 (75) | 0.25 (75) | 0.2 (60) |

Recruitment is planned to last 1 year and each participant is being followed for 1 year. To assess recruitment yields according to different targets, we stratify on ACEI/ARB and baseline  $\omega$ -3 use. The first stratum (people not using  $\omega$ -3) is randomized to placebo or  $\omega$ -3. The second stratum (people not using ACEI or ARB) is randomized to placebo or LO. The third stratum (people not using ACEI, ARB, or  $\omega$ -3) is randomized to placebo, LO, ω-3, or the combination. The original ENRGISE targets, based on the estimated proportions in LIFE are presented in Table 6.1. (We note that during the ENRGISE DSMB's August 23, 2016 phone call, the DSMB approved the investigators' request to lift the upper limit on the number recruited into stratum 1. In the text which follows, the original sample sizes remain as we do not know how many we will recruit into each stratum. The randomization weights will remain unchanged.) We expect to have a slight imbalance in the overall numbers within each treatment group of 90, 75, 75, and 60. Oversampling of the control group allows us to better estimate parameters associated with IL-6, walking speed, and major mobility disability in that group; this is important for planning the sample-size of the main trial. Note that anybody eligible for stratum 3 is also eligible for strata 1 and 2. To achieve overall balance between the two single interventions, we focus attention on having equal numbers in strata 1 and 2 but do not worry if either is less than 25% of the total as randomizing additional people in strata 3 provides similar information. If 20% were in each of strata 1 and 2, the overall weights would be 0.28, 0.24, 0.24, and 0.24; if 15%, then 0.26, 0.23, 0.23, and 0.28. Both are close to Table 6.1. and do not markedly reduce power for any comparison.

#### 6.2. Interventions and compliance. .

**6.2.a.** ω-3 fish oil and placebo (corn oil) are obtained by Epax in 0.7 g gel caps and they have identical shape, color, taste and weight. Each 0.7 g of fish oil ω-3 contains 400 mg eicosapentaenoic acid (EPA) and 200 mg docosahexaenoic acid (DHA). We start with 1.4 g/day of fish oil and continue until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not **decrease by ≥40%** vs. baseline (average of screening visits 1 and 2), we increase the dose to 2.8 g/day. To limit the effect of within subject variation, we use the average of 2 measures. If there is an acute illness within one month prior to the visit, the 3-month or the 6-month IL-6 measure is postponed or excluded from titration algorithms. In previous RCTs, ω-3 reduced IL-6 by >50% using 1 to 2 g/day of fish oil.<sup>75, 76</sup> In other trials in elders, fish oil was used in comparable doses

ranging from 0.6 to 2.3 g/day.62

# 6.2.a.1. Risks and risk protection and dose adjustments related to administration of $\omega$ -3

There are no contraindications to the use of  $\omega$ -3 fish oil, except intolerance or allergy to fish oil.  $\omega$ -3 are considered very safe and produce only mild adverse effects involving gastrointestinal upset and fishy aftertaste. The FDA has affirming menhaden fish oil as **Generally Recognized As Safe (GRAS)** under 21 CFR 4 184.1472 provided that the daily intake of EPA and DHA combined do not exceed 3 g per person per day. http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?fr=184.1472 and http://www.fda.gov/Food/IngredientsPackagingLabeling/GRAS/SCOGS/default.htm accessed on 9/11/2014.

 $\omega$ -3 may rarely cause clinical or subclinical bleeding, worsening of glycemic control in people with impaired glucose tolerance, rise in LDL cholesterol, and possibly hypotension when combined with antihypertensive treatment.

We start with a dose of 1.4 g/day of  $\omega$ -3 fish oil. Adverse effects, such as gastrointestinal discomfort are monitored. Dose will be adjusted as below based on serum glucose, LDL cholesterol and hemoglobin measured at baseline and at month 3, 6, and 9.  $\omega$ -3 fish oil dose will be decreased or discontinued if any of the following criteria are met at follow-up:

- New onset paroxysmal or persistent atrial fibrillation
- Hemoglobin decreases by ≥20% from baseline (dose will be discontinued),
- The participant is not diabetic and fasting glucose is > 126 AND has increased by >30% from baseline,
- The participant is diabetic and fasting glucose > 300,
- Baseline LDL > 130 AND increases by ≥ 20% from baseline,
- The participant is taking a blood pressure lowering agent OR is also participating in the Losartan arm of the study AND blood pressure is <90/50, or
- Participant does not tolerate the fish oil.

The principal investigator/study physician at each site has the discretion to opt out of  $\omega$ -3 fish oil dose adjustments due to glucose and/or LDL levels.

We increase the dose of  $\omega$ -3 fish oil to 2.8 g/day if the average of IL-6 measured at 3- and 6-month visits has not <u>decreased by at least 40%</u> vs. baseline (average of screening visits 1 and 2). The 40% threshold is selected based on previous trials with  $\omega$ -3 fatty acids.  $\omega$ -3 fatty acids have been shown to reduce IL-6 by >50% in RCTs<sup>75, 76</sup> and to be consistent with the threshold used below for losartan. To minimize the impact of outliers due to acute illness, the 3-month or the 6-month IL-6 measure are excluded or postponed if there is an acute illness within one month prior to the visit. In the rationale for dose titration we use the following assumptions:

- 1. IL-6 biovariation as a CV is ~30%. This is a reasonable estimate based on our own estimates (unpublished data) and those of others. <sup>150, 151</sup> This means that a SD of each person's day to day variability is about 30% of the mean value.
- 2. We have two measures at baseline that can be averaged to yield a reasonable estimate of each person's average value.
- 3. For dose adjustment we use IL-6 measured at 3 months and 6 months.
- 4. The half-life of IL-6 is extremely short (<30 minutes), so response to interventions is essentially coincident to the effect of the interventions.
- 5. We screen for outliers by excluding participants who experienced an acute illness within a month of the visit

**6.2.b.** LO and placebo (cellulose based) are obtained in 25 mg and 50 mg capsules. The shell capsules are cellulose based. Placebo and LO have identical shape, color, taste and weight. We start with 25 mg/day, if tolerated, we step up to 50 mg/day. If there are no safety concerns, we continue with 50 mg/day until the 6 month visit. If the average of IL-6 measured at 3- and 6-month visits does not **decrease by ≥40%** vs. baseline (average of screening visits 1 and 2), we increase the dose to 100 mg/day. Equivalent doses of ARBs have shown to reduce IL-6 by >40%<sup>77, 78</sup> and by 58%<sup>79</sup> in RCTs.

6.2.b.1. Risks, risk protection and dose adjustment related to administration of the ARB Losartan.

ARBs are reported to have a side effect profile indistinguishable from that of placebo but adverse reactions can occur rarely. Losartan has been safely used in large long-term clinical trials in older persons with congestive heart failure.<sup>83, 84</sup> ARBs are particularly well tolerated with very few side effects. Because ARBs do not influence kinin metabolism, dry cough is not seen and angioedema is very rare. Impairment in renal function may arise in patients with bilateral renal artery stenosis. Renal failure, reversible on discontinuation of ARB, may be precipitated.

- Hyperkalemia due to potassium retention mediated by reduction of aldosterone. Rare except in renal impairment.
- Impairment of renal function. Caution if bilateral renal artery stenosis suspected.
- Dizziness and syncope. Rare but may be precipitated by volume depletion.
- Angioedema. Very rare.
- Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) Including Selective Cyclooxygenase-2 Inhibitors
  (COX-2 Inhibitors): In patients who are elderly, volume-depleted (including those on diuretic therapy), or
  with compromised renal function, co-administration of NSAIDs, including selective COX-2 inhibitors,
  with angiotensin II receptor antagonists (including losartan) may result in deterioration of renal function,
  including possible acute renal failure. These effects are usually reversible. We monitor renal function
  periodically in patients receiving losartan and NSAID therapy as outlined below.

A full list of potential side effects of losartan can be found in the current package insert.

**6.3. Safety dose titration.** ARBs produce blood pressure reductions similar to those seen with ACE inhibitors and other antihypertensive classes. These drugs vary in efficacy and duration of action but all are recommended for once daily dosing. Like ACE inhibitors, duration of antihypertensive effects is dose-dependent; therefore, smooth blood pressure control over 24 hours is most likely at the maximum recommended dose. To avoid precipitous initial fall in blood pressure or decline in renal function, we start therapy with the lower dose of losartan (25 mg/day). If there are no safety concerns, the dose is increased to 50 mg/day and safety is again checked in about 1 week. To identify abrupt reduction in renal function that warrants drug dose reduction and to avoid dangerous hyperkalemia, we measure eGFR, potassium, and blood pressure before and soon (approximately 1 week) after starting losartan and after any dose adjustment. However, dose adjustments downward that are not related to renal function or hyperkalemia will not require a short-term follow-up blood draw.

In general, losartan dose will be maintained if ALL of the following criteria are met:

- Blood pressure is ≥ 100/50 and < 110/50,
- Potassium < 5.5,</li>
- eGFR has NOT declined by ≥ 20% from baseline, and
- No symptoms of lightheadedness or dizziness.

Losartan dose will be decreased if ALL of the following criteria are met:

- Blood pressure is ≥ 90/50 and < 100/50,</li>
- Potassium < 5.5,</li>
- eGFR has NOT declined by ≥ 20% from baseline, and
- · No symptoms of lightheadedness or dizziness.

Losartan dose will be stopped if ANY of the following criteria are met:

- Blood pressure < 90/50,</li>
- Potassium ≥ 5.5.
- eGFR decline ≥ 20% from baseline, or
- Symptoms of dizziness, lightheadedness, or syncope.

The principal investigator/study physician at each site has discretion to alter the losartan titration schedule on a case by case basis.

We increase the dose of losartan to 100 mg/day if the average of IL-6 measured at 3- and 6-month visits is not **decreased by at least 40%** vs. baseline (average of screening visits 1 and 2). The 40% threshold

was selected based on previous trials with ARBs. ARBs have been shown to <u>reduce IL-6 by >40%<sup>77, 78</sup> and by 58%<sup>79</sup> in RCTs</u>, and to be consistent with the threshold used above for  $\omega$ -3 fish oil. To minimize the impact of outliers due to acute illness, the 3-month or the 6-month IL-6 measure are excluded or postponed if there is acute illness within one month prior to the visit.

As part of the safety monitoring of the ENRGISE interventions, we measure blood pressure, blood hemoglobin, serum glucose, eGFR, LDL cholesterol, and potassium at baseline and at 3, 6, and 9 months of follow-up. In addition for those in the losartan arm of the trial, blood pressure, serum potassium, and eGFR, are measured about 1 week after randomization and about 1 week after any losartan dosage adjustment. However, serum potassium and eGFR are not measured one week after a downward dose adjustment that was not based on potassium or eGFR values.

**6.4. The Investigational New Drug (IND)** Per requirement of the Institutional Review Board, #IND124103 was submitted and approved by the FDA with the mention "STUDY MAY PROCEED"

## 6.5. Compliance

<u>To measure compliance</u> with LO and ω-3, we use dual methods involving both pill count<sup>152</sup> and participant recall. Pills are counted at each study visit.

# **6.6. Recruitment – inclusion/ exclusion criteria - (details in Table 6.2.)**

We identify men and women aged ≥70 years who are <u>able to complete the 400 m walk</u> at baseline, and are at <u>high risk of mobility disability</u> assessed by

- Self-reported difficulty walking ¼ mile or climbing a flight of stairs,
- <u>Usual walking speed <1 m/sec</u> and >0.44 m/sec on the 4 m walk (in the pilot phase we explore the feasibility of recruiting at least 50% of participants who have a baseline walking speed of <0.80 m/sec and >0.44 m/sec).<sup>22, 154, 155</sup> and
- <u>Chronic low-grade inflammation</u> measured by IL-6 >2.5 pg/ml, the threshold we have found for increased risk of mobility limitation, <sup>1, 2</sup> and <30 pg/ml to exclude high grade inflammation. To minimize within person variability, <sup>150, 156</sup> IL-6 is the average of 2 measures taken at screening visits, with the first measure being >2.3 and <30 pg/ml, and the average of the two measures >2.5 and <30 pg/ml.

We exclude subjects with acute, autoimmune and HIV illnesses and causes of low walking speed that may be related to neurological conditions, severe arthritis, or low vitamin D. Other exclusion criteria reflect conditions that may interfere with the conduct of the study, interventions or assessments. Those taking ACEI or ARB are excluded from the LO randomization and those eating>2 servings/week of fish in the past year or taking fish oil are excluded from the  $\omega$ -3 randomization. We recruit from the community. We use recruitment strategies successfully applied in LIFE, <sup>157</sup> LIFE-Pilot, <sup>158</sup> and TTrial, <sup>159</sup> which include primarily mass mailing, and newspaper, radio and TV ads and explore alternative recruitment strategies, such as electronic medical records to identify patients not taking study drugs and assess whether that strategy is effective in lieu of or in addition to mass mailing.

#### Table 6.2. Inclusion and exclusion criteria

#### **Inclusion Criteria**

- Men and women age ≥70 years
- Self-reported difficulty walking ¼ of a mile or climbing a flight of stairs
- Walking speed <1 m/sec and >0.44 m/sec on the 4 m walk at usual pace. A walking speed of <0.44 m/sec would not be compatible with completing the 400 m walk in 15 min. (In the pilot phase we explore the feasibility of recruiting at least 50% of participants who have a baseline walking speed of <0.80 m/sec and >0.44 m/sec)
- Able to complete the 400 m walk test within 15 minutes without sitting or the help of another person and without a walker, a
  cane is allowed
- Blood level IL-6 >2.5 pg/ml and <30 pg/ml.</li>
- Willingness to be randomized to the intervention groups

#### **Exclusion criteria**

- Failure or inability to provide informed consent
- Lives in a nursing home; persons living in assisted or independent housing are not excluded
- Self-reported inability to walk one block

- Significant cognitive impairment, defined as a known diagnosis of dementia, or a Mini-Mental State Exam (MMSE) score <24 (<23 for racial/ethnic minorities or participants with less than 9 years of education)
- Unable to communicate because of severe hearing loss or speech disorder
- Neurological conditions that are causing impaired muscle function or mobility (may include stroke with residual paresis, paralysis, neuropathy, Parkinson disease, or multiple sclerosis)
- Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, known active inflammatory or autoimmune disease (e.g. rheumatoid arthritis, lupus, Crohn's disease, HIV)
- Terminal illness with life expectancy less than 12 months
- Severe pulmonary disease, requiring either steroid pills or injections
- Other significant co-morbid disease that in the opinion of the field center PI would impair ability to participate in the trial, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar, schizophrenia), excessive alcohol use (>14 drinks per week); drug addiction; treatment for cancer (radiation or chemotherapy) within the past 1 year; or other conditions
- Lives outside of the study site or is planning to move out of the area in next 1 year or leave the area for >3 months during the
  next year
- Exclusion criteria that apply only to those who receive losartan:
  - Intolerance or allergy to ARBs
  - Known bilateral renal artery stenosis or liver cirrhosis
  - o Hypotension SBP<110 or DBP<60 mmHq
  - Serum potassium ≥5.0 mEq/L
  - Use of lithium salts
  - o eGFR < 15
  - Congestive heart failure with ejection fraction < 40%</li>
- Exclusion criteria that apply only to those who receive ω-3:
  - $\circ$  Intolerance or allergy to ω-3 or fish/shellfish
  - Fatty fish intake >2 servings per week on average
  - History of paroxysmal or persistent atrial fibrillation
- To maintain blinding, those who are not eligible to receive any active treatment (ω-3 or losartan) are excluded

#### Temporary exclusion criteria

- Myocardial infarction, CABG, or valve replacement within past 6 months;
- Pulmonary embolism or deep venous thrombosis within past 6 months;
- Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions;
- Stroke, hip fracture, hip or knee replacement, or spinal surgery within past 4 months;
- Physical therapy for gait, balance, or other lower extremity training within the past 2 months;
- Severe hypertension, e.g., SBP > 200, or DBP > 110 mmHg;
- Hemoglobin <10 g/dL
- Participation in another intervention trial within 3 months; participation in an observational study may be permitted;
- Current smoking (within 6 months),
- Acute infection (urinary, respiratory, other) or hospitalization within 1 month
- Exclusion criteria that apply only to those who receive losartan:
  - o Use of ACEI, ARB within 2 months
  - Use of aliskiren within 2 months in patients with type 2 diabetes or renal impairment with eGFR<60 <sup>161</sup>
  - Use of potassium sparing diuretics, other medications with potassium sparing properties (such as but not limited to spironolactone or eplerenone), potassium supplements, and salt substitutes containing potassium within 1 week
  - Transaminases >twice upper limit of normal to exclude participants with impaired liver function
- Exclusion criteria that apply only to those who receive ω-3:
  - $\circ$  Use of  $\omega$ -3 within 2 months

To maintain blinding, those who are not eligible to receive any active treatment ( $\omega$ -3 or losartan) are excluded

## 6.7. Outcomes

#### 6.7.a. Primary Outcomes

<u>IL-6 and walking speed during the 400 m walk test</u> are the main outcomes of the pilot study as outlined below.

The 400 m walk test at usual pace is used. Major mobility disability (MMD), 443, 162 defined as inability to walk 1/4 mile or 400 m, is measured in the pilot study and is our preferred primary outcome for the main trial. MMD is of major public health significance. Ability to walk 1/4 mile is measured in the US census 163 and in most epidemiologic surveys. The MMD outcome based on the 400 m walk test is a feasible, objective, reliable, 164 well-validated and important clinical and public health outcome in older people, 22, 143, 162 which has been

successfully implemented in the LIFE-Pilot and LIFE. 165, 166 We have shown it to be a more efficient outcome for clinical trials than self-reported disability or the Short Physical Performance Battery (SPPB). 167 Public health agencies use ability to walk ½ mile or 400 m to define need and policy impact of interventions. 18 Finally, people reporting the inability to walk 400 m incur higher health care costs of \$4,000 per person per year, compared with those not reporting inability to walk 400 m. 18-22 MMD is operationalized as the inability to complete a 400 m walk test within 15 min without sitting or help of another person or walker. 162 Completing the walk in >15 min would be in an extremely slow pace (<0.45 m/sec), which is of little utility in daily life. 168 A higher cut point (30 or 60 min), makes the assessment impractical and does not add to the clinical significance of the outcome. The time to walk 400 meters and the ability to complete the test provide data to test effects of the interventions resulting from both attenuation of decline and increase in walking speed. We hypothesize that the interventions reduce the risk of reaching the MMD outcome.

Non-completion of this test can be addressed by <u>adjudicating MMD</u> based on objective inability to walk 4 m in<a href="mailto:10">10</a> sec, or self- or proxy-reported inability to walk across a room.

# 6.7.b. Secondary and exploratory outcomes and measures

<u>SPPB.</u> A low score on the SPPB based on 4 m walk, balance & chair stands tests is a risk factor for disability, institutionalization, morbidity and mortality in initially non-disabled older persons.<sup>1-3</sup> The summary score and components of the SPPB have good reliability (ICCs range from 0.88 to 0.92).<sup>4,5</sup>

**Frailty** is a state of increased vulnerability to endogenous and exogenous stressors. <sup>169, 170</sup> Frailty involves fatigue, weight loss, infections, balance, strength and gait impairment leading to an increased risk of falls, delirium, and disability. In addition frailty is associated with inflammation <sup>43</sup> and thus it may be averted by anti-inflammatory interventions. We characterize frailty with Fried criteria developed by Fried et al. that employ self-reported exhaustion, unintentional weight loss, low energy expenditure, slow gait speed, and weak grip strength. <sup>171</sup> Those with >3 of the 5 factors are judged to be frail, those with 1 or 2 factors as pre-frail, and those

Isometric hand grip strength is a commonly used measure of upper body skeletal muscle function and has been widely used as a general indicator of functional status.  $^{172, 173}$  Higher IL-6 levels are associated with lower grip strength.  $^{3, 7, 174}$  Thus, reducing IL-6 with LO and ω-3 may result is higher grip strength vs. placebo. Grip strength in both hands is measured as we have successfully applied in LIFE.  $^{162}$ 

with no factors as non-frail.

# <u>Isokinetic dynamometry of the knee extensors and flexors.</u>

Participants complete this measure at baseline and 12 months. Observational studies have shown associations between knee extension isokinetic strength and physical functioning, disability and mortality.<sup>176</sup> The reliability of this

| Table 6.3. Schedule of screening, assessments and follow-up procedures in the pilot trial | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit type | Phone scr. | Scr. visit 1 | Scr. visit 2 | Base. Visit | Safety* | 3-Mo visit | Safety * | 6-Mo visit | Safety* | 9-Mo visit | Safety* | 12-Mo visit | Safety* | Extra visit** |
| Basic eligibility screening | | | | | | | | | | | | | | |
| Short consent and 4 m walk test | | Х | | | | | | | | | | | | |
| IL-6 | | Х | Х | | | x <sup>&amp;</sup> | | x <sup>&amp;</sup> | | x <sup>&amp;</sup> | | X <sup>&amp;</sup> | | |
| Medical history | | | Х | | | | | | | | | | | |
| MMSE | | | Х | | | | | | | | | | | |
| Safety blood tests | | | Х | Х | Х | Х | Х* | Х | Х* | Х | Х* | | Х* | Х |
| Additional biomarkers | | | | Х | | Х | | Х | | | | Х | | |
| Vital signs | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Anthropometric measures | | | | Х | | Х | | Х | | Х | | Х | | |
| Main Informed consent | | | | Х | | | | | | | | | | |
| Physical performance measures | | | Х | Х | | Х | | Х | | Х | | Х | | |
| Medical history update & adverse events | | | | Х | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Х | Х |
| Questionnaires | | | | Χ | | | | | | | | Χ | | |
| Dispense study drugs | | | | Χ | | Χ | | Χ | | Х | | | | |
| Assess compliance | | | | | | Х | | Х | | Х | | Х | | |
| Proxy interview (if needed) | | | | | | Х | | х | | Х | | Х | | |
| * DD and sorum notaceium and aCED are | | | ما سا | 4 | 4 | -1 | C4 41 | 1 4 | <b>∩</b> -l- | | 4:4 | | L | |

\* BP, and serum potassium and eGFR are measured about 1 week after the LO dose adjustment (potassium and eGFR are not measured if LO dose is reduced only for BP values). \*\* Extra visits if there are safety concerns. \* The IL-6 measure is excluded or postponed if there has been an acute illness within one month prior to the visit

measure is generally excellent.<sup>177, 178</sup> In addition, several randomized trials in older mobility limited populations have shown this measure to be responsive to therapeutic interventions.<sup>179, 180</sup>

The Short Form (SF-36) Health Survey 181-184 is administered to assess the general health status as

Participant Reported Outcomes (PRO).

## 6.8. Screening, assessments and follow-up (Table 6.3.)

Potential participants are screened by telephone interviews to assess the main inclusion/exclusion criteria. Those who qualify are invited for the first screening visit during which a brief informed consent is obtained and the 4 m walk at usual pace is administered. Blood level of IL-6 is tested in those with a walking speed <1 m/sec and >0.44 m/sec. Participants with qualifying IL-6 levels are invited for the second screening visit to review medical history and current medications, complete blood testing (vitamin D, CBC, chemical panel, and second IL-6 measure), vital signs (blood pressure, pulse and temperature), 400 m walk, and the Mini Mental State Examination (MMSE). 185 The study medical safety officer will review the participant's health history, medication use, vital signs, and laboratory test results, and clear for randomization according to the study inclusion and exclusion criteria. If there are no safety concerns, participants attend the baseline visit during which the following is completed: full informed consent, questions to assess frailty, 171 blood collection for labs, vital signs and anthropometric measurements, the SPPB, isokinetic dynamometry of the knee extensors and flexors, grip strength, and questionnaires. Validated Minnesota physical activity<sup>186</sup>, depressive symptoms (CES-D)<sup>175</sup>, patient reported outcomes (SF-36), and fatigability<sup>198</sup> questionnaires are completed at the baseline and 12 month visit. The physical activity results are used as potential modifiers in the data analyses. If there are no exclusion criteria identified, the participants are randomized, and the study drugs are dispensed. The baseline measures are repeated as outlined in Table 6.3. BP&P, blood tests and adverse events are measured about 1 week after randomization and after each visit when the LO dose is modified. Medication dose is adjusted as outlined in the above titration and safety algorithms.

- **6.9. Measure of additional biomarkers** Inflammation, characterized by higher blood cytokine levels related to the activation of innate immunity and other systems (coagulation), is part of the aging process, plays a role in virtually all diseases, and contributes to mobility limitations. While it is known that inflammation markers predict these outcomes and mortality, little is known about how anti-inflammatory interventions affect the plasma cytokine levels, or associated pathways. Thus, we measure novel and established markers of inflammation and aging at baseline, and follow-up, and relate these to both change in IL-6 and change in walking speed to:
- (1) Characterize the effect of the interventions on these cytokines: (1.a.) Are these cytokines/pathways impacted by the interventions? (1.b) Are the changes in these markers pre- vs. post-intervention less than, equivalent to, or greater than that of IL-6?
- (2) Assess if these biomarkers yield independent information from IL-6 with respect to the change in walking speed and/or provide benefit for screening participants in the main ENRGISE trial.

# 6.10 Data analyses and power for the ENRGISE Pilot Study and biomarkers assays

The data analyses and power section is presented in the order by which the aims are likely to be achieved rather than the order in which the aims are stated elsewhere in the protocol.

#### 6.10.a. Feasibility and recruitment

Feasibility of recruitment and identifying the study population are contained in Aim a (ii). In the ENRGISE Pilot Study we will use one-sided tests/confidence intervals because we wish to rule out conditions that would make the main study infeasible. Having a higher than hypothesized safe tolerable rate, higher yield for recruitment, or stronger relationship between the changes in IL-6 and walking speed would simply make the follow-up study easier to implement. For efficacy, we use tests at the 10% significance level;<sup>187, 188</sup> this is consistent with the FDA's aims for phase 2 versus phase 3 studies.<sup>189, 190</sup> No formal adjustment for multiple comparisons is planned for the pilot study.

We assess the recruitment yields in strata 1-3 presented in Table 6.1 and the proportions of people who tolerate LO and  $\omega$ -3. One-sided exact confidence intervals of these proportions are calculated. If we need to screen 300 people to recruit 75 into strata 1 (People not using  $\omega$ -3) or 2 (People not using ACEI or ARB) (25% yield), the 95% one-sided CI would set the lower bound of our recruitment yield at 20.9% using a Clopper-Pearson interval<sup>191</sup> and 8.3% if we need to screen 750 (10% yield). For stratum 3 (People not using ACEI, ARB, or  $\omega$ -3) (target 150), these lower limits would be 22.1% (25% yield) or 8.8% (10% yield). Note that those eligible for stratum 3 are also eligible for strata 1 and 2; these people are also used to estimate the

proportions eligible; thus, our CIs above are conservative.

#### 6.10.b. Intervention Effect

We use the "intention to treat" approach assuming participants are grouped according to randomization for all analyses of the intervention effect. The stratified recruitment and randomization allow us to compare mean log(IL-6) between each of the three active groups to placebo using a linear mixed model with both main effects and their interaction, adjusted for baseline log(IL-6) and strata. Time is a repeated factor, and the primary comparison is based on a contrast at 12 months. The covariance structure will be assumed to be unstructured. The primary focus is on marginal comparisons (135 and 165/group) between each active intervention and placebo using one-sided hypothesis tests at the 10% level (we are not looking for definitive evidence, but to rule out small effects). We assume 5% loss to follow-up (LTFU); this is similar to the 5% we achieved in LIFE. Using the root mean squared error from LIFE-P (adjusted for baseline log(IL-6) and treatment) of 0.52, we have 91% power to detect a difference if the difference (on the log scale) is at least 0.1625. This is equivalent to the difference between 4.20 and 3.57 pg/ml (or a 15% difference). We would have 66% power for a 10% difference (4.20 vs. 3.78 pg/ml, 0.1054 on the log scale) and 99% power for a 20% difference (4.20 vs. 3.36 pg/ml, 0.2231 on the log scale). Individual treatment group comparisons (at least 60 vs. 75/group) would have 44% power for a 10% difference, 68% power for a 15% difference, and 87% power for a 20% difference. This achieves the first part of Aim a (i). As sensitivity analyses, we also explore the impact of additional factors (e.g., diet, physical activity, medication use) by adding these factors to the models. Although the mixed model is robust against data missing at random (MAR), multiple imputation will be used in sensitivity analyses.

From LIFE-Pilot, the SD of 400 m walk speed in IL-6 eligible participants is 0.21 m/s, with high correlation (r>0.80) between baseline and 12 month measures. With at least 60 and 75 participants per group (for pairwise comparisons), we project to have >99% power to detect a difference in means of >0.095 m/sec using a one-sided test at the 10% level (a substantial meaningful change). 192 There is also 67% power to detect a >0.038 m/sec difference (a small meaningful change). Using groups of 135 and 165 (for main effects), we would have >99% power to detect >0.095 m/sec, and 86% power for a difference >0.038 m/sec in walking speed. This analysis uses linear mixed models, as for IL-6; a similar approach is used for the secondary outcomes of SPPB, frailty, and grip strength. This achieves the last part of Aim a (i). For people who are unable to complete the 400m walk, we will use their walking speed from the portion completed.

## 6.10.c. Associations between inflammation and function

We base our calculation of detectable SPPB effects on LIFE data. The correlations between baseline and 24 month follow-up SPPB outcomes were 0.49 (Successful Aging: SA) and 0.47 (Physical Activity: PA); we assume a correlation of 0.5 between baseline and 12 month in ENRGISE. Estimated standard deviations at 24 months were 2.60 (SA) and 2.47 (PA); we assume 2.5. Under these assumptions, for the comparisons of 60 to 65 people, we have 90% power to detect a difference of at least 0.99 SPPB units; for the comparisons of 135 to 165 people, we have 90% power to detect a difference of at least 0.66 SPPB units. Both assume 1-sided tests at the 10% level.

We will examine the relationship between the change in IL-6 and the change in walking speed using univariate regression. Assuming we assess ≥285 participants (of 300, ≥95%) at 12 months, we have 80% power to detect a correlation less than -0.126 (i.e. at least 1.59% of explained variability) using a one-sided test at the 10% level. We have 90% power if the correlation is less than -0.152 (Aim a (iii)).

To assess intra-person variability in IL-6 (Aim a (iii)), we measure IL-6 at both screening visits. We use a Bland-Altman plot to assess agreement; this is summarized using a 95% CI of the difference at the two visits providing information on the expected differences over one week due to biological variability and measurement error. If agreement is high, one measure is likely sufficient for recruitment into the main study. If not, we may need to use two or more measures to determine eligibility and to assess participant-specific risk.

#### 6.10.d. Additional inflammatory biomarkers:

In addition to IL-6 levels, we examine additional markers of inflammation (Aim b (i) and (ii)). As with IL-6, our primary focus is on the relationships between changes in cytokines with the change in walking speed using linear mixed models. We use stratified linear mixed models (as described above for IL-6) to examine the impact of interventions on these cytokines. These analyses assess whether changes in these cytokines are of similar magnitude to IL-6. As the absolute levels differ between cytokines, focus is on relative changes from baseline. We also examine these cytokines in models also including baseline and follow-up log(IL-6) to assess whether they provide additional predictive information. We also explore MMD event rates by baseline levels of IL-6 and additional cytokines to explore whether we can use an additional cytokine to select a population at greater risk to use for the main study, recognizing the potential tradeoff between ease of recruitment and selecting a population at higher risk.

# 6.10.e. Informing the main study

We assess compliance and retention rates (Aim a (ii)). Although we expect to be underpowered for incident mobility disability, we collect these data and compare estimates of event rates to those obtained in SA group LIFE participants that would have been eligible for ENRGISE (Aim a (ii)). While power is limited, we also examine whether there is sub-additivity and interaction of interventions in stratum 3, which supports the decision of whether to proceed with a factorial or parallel group design in Phase 3 (Aim a (ii)).

We integrate all available information to make a determination about which approaches to carry forward into the main study. Weighed in this decision is recruitment yield (is it practical to consider a full size trial?), safety and tolerability (do participants tolerate the interventions?), changes in IL-6 in the pilot studies, the relationship of change in IL-6 with change in walking speed, the conclusions from our data analysis of other studies (e.g. LIFE, Look AHEAD, Health ABC, CLIP), and a revised literature search. Finally, we combine all information to estimate the sample size and **cost of the main trial** (Aim a (ii)). For example, for a two-arm study, we would need 2,084 people to have 90% power to detect a 20% (HR=0.8) reduction in MMD assuming a two-sided test at the 5% level, a control group event rate of 18.3%/year, LTFU of 5%/year, 18 months of recruitment, and a total study length of 4 years. To detect a 25% effect (HR=0.75), we would need 1,296 people. These calculations use the estimated MMD rate of 18.3%/year in the control group among people in LIFE-P whose baseline IL-6 was between 2.5 and 10 pg/ml.

## 7. Possible Discomforts and Risks

# 7.1. Confidentiality

Lack of maintenance of confidentiality is a potential risk. The information below relates to all collaborating performance sites for the proposed study. Data are used only in aggregate and no identifying characteristics of individuals will be published or presented. Results of testing are sent to participant's private physicians if participants agree to this. Alert values for medically relevant procedures (e.g., blood pressure, pulse rate, MMSE, blood tests) are sent to participants and participants' physicians, depending on the urgency of the values.

Confidentiality of data is maintained by using research identification numbers that uniquely identify each individual. Safeguards are established to ensure the security and privacy of participants' study records. Appropriate measures are taken to prevent unauthorized use of study information. The research ID number is used. The research records are kept in a locked room in the Field Center. The files matching participants' names and demographic information with research ID numbers are kept in a locked file. Only trained and certified study personnel has access to these files. After the study is completed, local data are stored with other completed research studies in a secured storage area.

In compliance with the Health Insurance Portability and Accountability Act (**HIPAA**) and the Standards for Privacy of Individually Identifiable Health Information of the Department of Health and Human Services, we access personal health information and medical records only after receiving signed informed consent.

## 7.2. Biological samples repository

We comply with the Office of Extramural Research requirements and guidelines related to the research use of stored biological specimens. The repository is subject to the oversight of the University of Vermont IRB which reviews and approves the protocol, training documents, and an informed consent document, according to the elements described above, for distribution to collector-investigators and their local IRBs.

# 7.3. Safety, risks, risk protection and dose adjustment related to drug administration is discussed above in section 6.

## 7.4. Safety measures during the assessments

All study assessments are done by staff trained and certified in Good Clinical Practice, study procedures and assessments, and safety procedures. The study nurse/medical safety officer reviews all health assessments, vital signs, medical history, medication use, and blood tests. All assessors receive **CPR training** and training on management of acute events including syncope, chest pain, acute dyspnea and abnormal vital signs. All sites have on-call access to contact numbers for emergency services.

**Phlebotomy.** The risks of drawing blood from a vein or finger stick include discomfort at the site of puncture; possible bruising and swelling around the puncture site; rarely an infection; and, uncommonly, faintness from the procedure.

**Blood pressure measurement.** The risks of placing a blood pressure cuff on a participant's arms are that it may cause pinching or slight bruising.

**400 m walk test.** The 400 m walk test may be associated with the risk of falling or development of chest discomfort due to coronary ischemia or dyspnea due to heart failure or lung disease. Rarely, falling during the 400 m walk test may result in a fracture.

Research staff members that collect data are trained and certified in 400 m walk testing before they work with study participants. Study staff members are trained not to administer the 400 m walk test if they feel or the participant feels that testing is unsafe. Safety precautions are taken during the 400 m walk test by applying standardized stopping criteria. If the participant reports pain, tightness or pressure in the chest, significant shortness of breath, feeling faint, lightheaded or dizzy, or significant other medical problems the test is stopped. In addition, participants are asked whether they feel the test is safe. Those who state it may be unsafe are not allowed to complete the test. Staff members are trained to protect against falling and are trained in CPR. They are trained in activating the local emergency response system. In our experience conducting thousands of 400 m walk tests on individuals within various studies, the risk of falling is less than 1/500 and the risk of a fracture-associated fall is less than 1/5000.

In the LIFE study we have performed approximately 10,000 400 m walk tests with no safety concerns raised by the DSMB.

**SPPB assessment.** Similar to the **400 m** walk test, completion of the SPPB may be associated with the risk of falling or development of chest discomfort due to coronary ischemia or dyspnea due to heart failure or lung disease. Rarely, falling during the SPPB test may result in a fracture. Research staff members who collect data are trained and certified in SPPB measurement.

**Strength measures**, may rarely cause pain or muscle sprain. In our experience conducting thousands of measures, the testing has demonstrated to be safe.

#### Questionnaire administration.

Participation includes a risk of loss of confidentiality of personal health information. A number of methods are employed to maintain confidentiality of participants. First, questionnaire data are collected in secure spaces where the interview cannot be overheard. Secondly, only study investigators and key research staff (i.e. study

programmers and biostatisticians) have access to the study database. Third, participants are assigned a unique study identifier. Individual names are removed from the study database and only the unique study identifier is used to distinguish participants in the database. Fourth, collected data are maintained in locked computer files and file cabinets to which only study investigators have access. Collected data are used only for research purposes. Published data will not contain any individual identifiers.

## Participant burden and fatigue

The duration of clinic visits for screening, baseline, and follow-up range between <u>15 min to 3 hours</u>. If a participant becomes too fatigued we make arrangements for a second visit or to complete the testing in the participant's home. Based on our experience with LIFE-Pilot, LIFE and other RCTs in the elderly (SHEP), with observational studies in healthy older persons (CHS<sup>195</sup> and Health ABC<sup>196</sup>), and with disabled elderly women (WHAS), visits lasting between 2 and 4 hours did not negatively affect annual follow-up **retention**, which was >90%. We closely **monitor** the potential impact of visit burden on retention. This information will be used to promptly implement strategies to promote retention and adherence.

# 7.5. Data Safety and Monitoring Plan

## Monitoring adverse events

**Safety** of the study participants is always our major concern. The **Intervention and Safety Committee** provides early monitoring of adverse events and ensures standardization of clinical practice and safety issues across all sites.

An **adverse event** is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

The event is **serious** if it results in death, is life-threatening, requires inpatient hospitalization or prolongs an existing hospitalization, results in a persistent or significant disability/incapacity, or congenital anomaly/birth defect.

Safety related events are reported in a timely fashion, as required by the NIH, FDA, DSMB and the IRBs that are responsible for study oversight.

The classification of potential relationship to the intervention is as follows.

**Definite** Temporal pattern + Known or expected AE response pattern + Confirmed by

stopping the intervention + Reappearance of AE on re-challenge

Possible Temporal pattern + Known or expected AE response pattern + Could have been

produced by a number of other factors

**Not related** AE for which sufficient information exists to indicate that the cause is unrelated to

the study intervention

ENRGISE study participants are comprised of a frail, elderly population expected to be at high risk for acute and chronic comorbid health events.

A **Data and Safety Monitoring Plan (DSMP)** is implemented to ensure the safety of all participants involved in the study and to ensure the validity and integrity of the data. The Principal Investigators with the advice and assistance of the Intervention and Safety Committee described below and the Steering committee monitor all aspects of safety. The Intervention and Safety Committee reviews all Serious, Unexpected, and Onsite adverse events and makes recommendations to the Steering Committee for any changes in reporting, consent or study activities.

A **Data Safety Monitoring Board (DSMB)** is established, with responsibility to monitor all aspects of the study, including those that require access to any masked data. The DSMB and its chair are named and approved by the NIA. It is planned that the DSMB meets by conference call as determined by the DSMB and the NIA. The DSMB has access to all study data, documents and progress. The Intervention and Safety Committee, **comprised of safety personnel from each site, the Chair, and a representative of the DMAQC** reports to the DSMB for issues related to participant safety.

The DSMB has the following charges:

- Review the study protocol.
- Review data (including masked data) over the course of the trial.
- Identify problems relating to safety over the course of the study.
- Identify needs for additional data relevant to safety issues and request these data from the study investigators.
- Propose appropriate analyses and periodically review developing data on safety and endpoints.
- Make recommendations regarding recruitment, treatment effects, retention, compliance, safety issues and continuation of the study.
- At any time, the DSMB may recommend discontinuation of any component/treatment group of the study

Finally, the NIA makes the final decision on whether or not to accept the DSMB's recommendation about discontinuation of any component of the study. Any serious adverse event that might be due to the study intervention are reported to the DSMB, the IRBs, and to the NIA Project Office. The exact timeline for reporting serious adverse events is determined by the DSMB, IRBs, and NIA.

## 8. Potential benefits of the proposed research to subjects and to others

There is direct benefit to the study participants, including study blood tests and a comprehensive assessment of physical function. All study participants are encouraged to communicate the results from the study to their primary care providers.

ENRGISE will provide critical information regarding the efficacy of the study interventions in averting low-grade chronic inflammation and mobility impairments in vulnerable older adults. The results of ENRGISE will have relevant clinical and public health implications, and will fill an important gap in knowledge for practicing evidence-based geriatric medicine.

We believe that the aforementioned risks of this study are minimal and reasonable, when compared to 1) the scientific knowledge to be gained by performing these studies as well as 2) the potential benefits to study subjects.

#### 9. Conflict of Interest

None

#### Reference List

- 1. Penninx BW, Kritchevsky SB, Newman AB, Nicklas BJ, Simonsick EM, Rubin S, Nevitt M, Visser M, Harris T, Pahor M. Inflammatory markers and incident mobility limitation in the elderly. J Am Geriatr Soc 2004; 52(7):1105-1113.
- 2. Ferrucci L, Harris TB, Guralnik JM, Wacholder S, Tracy RP, Corti MC, Penninx BWJH, Pahor M, Wallace RB, Havlik RJ. Inflammation, a novel risk factor for disability in older persons. J Am Geriatr Soc 1999; 47:639-646.
- 3. Cesari M, Penninx BW, Pahor M, Lauretani F, Corsi AM, Guralnik JM, Ferrucci L. Inflammatory markers and physical performance in older persons: the InChianti study. J Gerontol A Biol Sci Med Sci 2004; 59:242-248.
- 4. Sanders JL, Ding V, Arnold AM, Kaplan RC, Cappola AR, Kizer JR, Boudreau RM, Cushman M, Newman AB. Do changes in circulating biomarkers track with each other and with functional changes in older adults? J Gerontol A Biol Sci Med Sci 2014; 69(2):174-181. PMCID: PMC4038245
- 5. Singh T, Newman AB. Inflammatory markers in population studies of aging. Ageing Res Rev 2011; 10(3):319-329. PMCID: PMC3098911
- 6. Hsu FC, Kritchevsky SB, Liu Y, Kanaya A, Newman AB, Perry SE, Visser M, Pahor M, Harris TB, Nicklas BJ. Association Between Inflammatory Components and Physical Function in the Health, Aging, and Body Composition Study: A Principal Component Analysis Approach. J Gerontol A Biol Sci Med Sci 2009; 64(5):581-589.
- 7. Brinkley TE, Leng X, Miller ME, Kitzman DW, Pahor M, Berry MJ, Marsh AP, Kritchevsky SB, Nicklas BJ. Chronic inflammation is associated with low physical function in older adults across multiple comorbidities. J Gerontol A Biol Sci Med Sci 2009; 64(4):455-461.
- 8. Penninx BW, Abbas H, Ambrosius W, Nicklas BJ, Davis C, Messier SP, Pahor M. Inflammatory Markers and Physical Function Among Older Adults with Knee Osteoarthritis. J Rheumatol 2004; 31(10):2027-2031.
- 9. Cesari M, Marzetti E, Laudisio A, Antonica L, Pahor M, Bernabei R, Zuccala G. Interaction of HDL cholesterol concentrations on the relationship between physical function and inflammation in community-dwelling older persons. Age Ageing 2010; 39(1):74-80.
- 10. McDermott MM, Liu K, Ferrucci L, Tian L, Guralnik JM, Green D, Tan J, Liao Y, Pearce WH, Schneider JR, McCue K, Ridker P, Rifai N, Criqui MH. Circulating blood markers and functional impairment in peripheral arterial disease. J Am Geriatr Soc 2008; 56(8):1504-1510. PMCID: PMC2658758
- 11. Verghese J, Holtzer R, Lipton RB, Wang C. High-sensitivity C-reactive protein and mobility disability in older adults. Age Ageing 2012; 41(4):541-545. PMCID: PMC3500856
- 12. Oh DY, Talukdar S, Bae EJ, Imamura T, Morinaga H, Fan W, Li P, Lu WJ, Watkins SM, Olefsky JM. GPR120 is an omega-3 fatty acid receptor mediating potent anti-inflammatory and insulin-sensitizing effects. Cell 2010; 142(5):687-698. PMCID: PMC2956412
- 13. Saltiel AR. Fishing out a sensor for anti-inflammatory oils. Cell 2010; 142(5):672-674.

- Benicky J, Sanchez-Lemus E, Pavel J, Saavedra JM. Anti-inflammatory effects of angiotensin receptor blockers in the brain and the periphery. Cell Mol Neurobiol 2009; 29(6-7):781-792. PMCID: PMC2718067
- 15. Feng X, Luo Z, Ma L, Ma S, Yang D, Zhao Z, Yan Z, He H, Cao T, Liu D, Zhu Z. Angiotensin II receptor blocker telmisartan enhances running endurance of skeletal muscle through activation of the PPAR-delta/AMPK pathway. J Cell Mol Med 2011; 15(7):1572-1581.
- 16. Shumway-Cook A, Patla A, Stewart A, Ferrucci L, Ciol MA, Guralnik JM. Environmental components of mobility disability in community-living older persons. J Am Geriatr Soc 2003; 51(3):393-398.
- 17. Shumway-Cook A, Patla AE, Stewart A, Ferrucci L, Ciol MA, Guralnik JM. Environmental demands associated with community mobility in older adults with and without mobility disabilities. Phys Ther 2002; 82(7):670-681.
- Hardy SE, Kang Y, Studenski SA, Degenholtz HB. Ability to walk 1/4 mile predicts subsequent disability, mortality, and health care costs. J Gen Intern Med 2011; 26(2):130-135. PMCID: PMC3019329
- 19. Hoffman JM, Ciol MA, Huynh M, Chan L. Estimating transition probabilities in mobility and total costs for medicare beneficiaries. Arch Phys Med Rehabil 2010; 91(12):1849-1855. PMCID: PMC3404130
- 20. Hardy SE, Perera S, Roumani YF, Chandler JM, Studenski SA. Improvement in usual gait speed predicts better survival in older adults. J Am Geriatr Soc 2007; 55(11):1727-1734.
- 21. Hoffman JM, Shumway-Cook A, Yorkston KM, Ciol MA, Dudgeon BJ, Chan L. Association of mobility limitations with health care satisfaction and use of preventive care: a survey of Medicare beneficiaries. Arch Phys Med Rehabil 2007; 88(5):583-588.
- 22. Newman AB, Simonsick EM, Naydeck EM, Kritchevsky SB, Nevitt M, Pahor M, Satterfield S, Brach JS, Studenski SA, Harris TB. Association of long-distance corridor walk performance with mortality, cardiovascular disease, mobility limitation, and disability. JAMA 2006; 295(17):2018-2026.
- 23. Giovannini S, Onder G, Liperoti R, Russo A, Carter C, Capoluongo E, Pahor M, Bernabei R, Landi F. Interleukin-6, C-Reactive Protein, and Tumor Necrosis Factor-Alpha as Predictors of Mortality in Frail, Community-Living Elderly Individuals. J Am Geriatr Soc 2011; 59(9):1679-1685.
- 24. Newman AB, Sachs MC, Arnold AM, Fried LP, Kronmal R, Cushman M, Psaty BM, Harris TB, Robbins JA, Burke GL, Kuller LH, Lumley T. Total and cause-specific mortality in the cardiovascular health study. J Gerontol A Biol Sci Med Sci 2009; 64(12):1251-1261. PMCID: PMC2773812
- 25. Harris TB, Ferrucci L, Tracy RP, Corti MC, Wacholder S, Ettinger WH, Jr., Heimovitz H, Cohen HJ, Wallace R. Associations of elevated interleukin-6 and C-reactive protein levels with mortality in the elderly. Am J Med 1999; 106(5):506-512.
- 26. Brinkley TE, Hsu FC, Beavers KM, Church TS, Goodpaster BH, Stafford RS, Pahor M, Kritchevsky SB, Nicklas BJ. Total and Abdominal Adiposity Are Associated With Inflammation in Older Adults Using a Factor Analysis Approach. J Gerontol A Biol Sci Med Sci 2012; 67(10):1099-1106. PMCID: PMC3437966
- 27. Campisi J, Andersen JK, Kapahi P, Melov S. Cellular senescence: a link between cancer and agerelated degenerative disease? Semin Cancer Biol 2011; 21(6):354-359. PMCID: PMC3230665

- 28. Roubenoff R. The "cytokine for gerontologists" has some company. J Gerontol A Biol Sci Med Sci 2014; 69(2):163-164.
- 29. Anand S, Johansen KL, Kurella TM. Aging and chronic kidney disease: the impact on physical function and cognition. J Gerontol A Biol Sci Med Sci 2014; 69(3):315-322. PMCID: PMC4017829
- 30. Folsom AR, Pankow JS, Tracy RP, Arnett DK, Peacock JM, Hong Y, Djousse L, Eckfeldt JH. Association of C-reactive protein with markers of prevalent atherosclerotic disease. Am J Cardiol 2001; 88(2):112-117.
- 31. Libby P, Sukhova G, Lee RT, Galis ZS. Cytokines regulate vascular functions related to stability of the atherosclerotic plaque. J Cardiovasc Pharmacol 1995; 25 Suppl 2:S9-12.
- 32. Ferrucci L, Penninx BW, Volpato S, Harris TB, Bandeen-Roche K, Balfour J, Leveille SG, Fried LP, Md JM. Change in muscle strength explains accelerated decline of physical function in older women with high interleukin-6 serum levels. J Am Geriatr Soc 2002; 50(12):1947-1954.
- 33. Schaap LA, Pluijm SM, Deeg DJ, Harris TB, Kritchevsky SB, Newman AB, Colbert LH, Pahor M, Rubin SM, Tylavsky FA, Visser M. Higher inflammatory marker levels in older persons: associations with 5-year change in muscle mass and muscle strength. J Gerontol A Biol Sci Med Sci 2009; 64(11):1183-1189.
- 34. Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Inflammation, aspirin, and the risk of cardiovascular disease in apparently healthy men. N Engl J Med 1997; 336:973-979.
- 35. Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Plasma concentration of C-reactive protein and risk of developing peripheral vascular disease. Circulation 1998; 97(5):425-428.
- 36. Ridker PM, Glynn RJ, Hennekens CH. C-reactive protein adds to the predictive value of total and HDL cholesterol in determining risk of first myocardial infarction. Circulation 1998; 97:2007-2011.
- 37. Cesari M, Penninx BWJH, Newman AB, Kritchevsky SB, Nicklas BJ, Sutton-Tyrrell K, Tracy RP, Rubin S, Harris TB, Pahor M. Inflammatory markers and cardiovascular disease (The Health, Aging and Body Composition [Health ABC] Study). Am J Cardiol 2003; 92:522-528.
- 38. Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM, Jr., Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med 2008; 359(21):2195-2207.
- 39. Ridker PM, Luscher TF. Anti-inflammatory therapies for cardiovascular disease. Eur Heart J 2014.
- 40. Everett BM, Pradhan AD, Solomon DH, Paynter N, Macfadyen J, Zaharris E, Gupta M, Clearfield M, Libby P, Hasan AA, Glynn RJ, Ridker PM. Rationale and design of the Cardiovascular Inflammation Reduction Trial: a test of the inflammatory hypothesis of atherothrombosis. Am Heart J 2013; 166(2):199-207. PMCID: PMC3888829
- 41. Ridker PM, Thuren T, Zalewski A, Libby P. Interleukin-1beta inhibition and the prevention of recurrent cardiovascular events: rationale and design of the Canakinumab Anti-inflammatory Thrombosis Outcomes Study (CANTOS). Am Heart J 2011; 162(4):597-605.
- 42. Goodman MN. Interleukin-6 induces skeletal muscle protein breakdown in rats. Proc Soc Exp Biol Med 1994; 205(2):182-185.

- 43. Walston J, McBurnie MA, Newman A, Tracy RP, Kop WJ, Hirsch CH, Gottdiener J, Fried LP. Frailty and activation of the inflammation and coagulation systems with and without clinical comorbidities: results from the Cardiovascular Health Study. Arch Intern Med 2002; 162(20):2333-2341.
- 44. Boxer RS, Dauser DA, Walsh SJ, Hager WD, Kenny AM. The association between vitamin D and inflammation with the 6-minute walk and frailty in patients with heart failure. J Am Geriatr Soc 2008; 56(3):454-461.
- 45. Nicklas BJ, Ambrosius W, Messier SP, Miller GD, Penninx BWJH, Loeser RF, Palla S, Bleecker GC, Pahor M. Dietary-induced weight loss, exercise and chronic inflammation in older, obese adults: A randomized controlled clinical trial. Am J Clin Nutr 2004; 79:544-551.
- 46. Nicklas BJ, Hsu FC, Brinkley TJ, Church T, Goodpaster BH, Kritchevsky SB, Pahor M. Exercise training and plasma C-reactive protein and interleukin-6 in elderly people. J Am Geriatr Soc 2008; 56(11):2045-2052. PMCID: PMC2683336
- 47. Li H, Malhotra S, Kumar A. Nuclear factor-kappa B signaling in skeletal muscle atrophy. J Mol Med (Berl) 2008; 86(10):1113-1126. PMCID: PMC2597184
- 48. Merritt EK, Stec MJ, Thalacker-Mercer A, Windham ST, Cross JM, Shelley DP, Craig TS, Kosek DJ, Kim JS, Bamman MM. Heightened muscle inflammation susceptibility may impair regenerative capacity in aging humans. J Appl Physiol (1985) 2013; 115(6):937-948. PMCID: PMC3764621
- 49. Youm YH, Grant RW, McCabe LR, Albarado DC, Nguyen KY, Ravussin A, Pistell P, Newman S, Carter R, Laque A, Munzberg H, Rosen CJ, Ingram DK, Salbaum JM, Dixit VD. Canonical Nlrp3 inflammasome links systemic low-grade inflammation to functional decline in aging. Cell Metab 2013; 18(4):519-532. PMCID: PMC4017327
- 50. Toth MJ, Matthews DE, Tracy RP, Previs MJ. Age-related differences in skeletal muscle protein synthesis: relation to markers of immune activation. Am J Physiol Endocrinol Metab 2005; 288(5):E883-E891.
- 51. Srivastava AK, Qin X, Wedhas N, Arnush M, Linkhart TA, Chadwick RB, Kumar A. Tumor necrosis factor-alpha augments matrix metalloproteinase-9 production in skeletal muscle cells through the activation of transforming growth factor-beta-activated kinase 1 (TAK1)-dependent signaling pathway. J Biol Chem 2007; 282(48):35113-35124.
- 52. Phillips T, Leeuwenburgh C. Muscle fiber specific apoptosis and TNF-alpha signaling in sarcopenia are attenuated by life-long calorie restriction. FASEB J 2005; 19(6):668-70.
- 53. Tchkonia T, Zhu Y, van DJ, Campisi J, Kirkland JL. Cellular senescence and the senescent secretory phenotype: therapeutic opportunities. J Clin Invest 2013; 123(3):966-972. PMCID: PMC3582125
- 54. Calvani R, Joseph AM, Adhihetty PJ, Miccheli A, Bossola M, Leeuwenburgh C, Bernabei R, Marzetti E. Mitochondrial pathways in sarcopenia of aging and disuse muscle atrophy. Biol Chem 2013; 394(3):393-414. PMCID: PMC3976204
- 55. Lucas L, Russell A, Keast R. Molecular mechanisms of inflammation. Anti-inflammatory benefits of virgin olive oil and the phenolic compound oleocanthal. Curr Pharm Des 2011; 17(8):754-768.
- 56. Oh dY, Walenta E, Akiyama TE, Lagakos WS, Lackey D, Pessentheiner AR, Sasik R, Hah N, Chi TJ, Cox JM, Powels MA, Di SJ, Sinz C, Watkins SM, Armando AM, Chung H, Evans RM, Quehenberger O,

- McNelis J, Bogner-Strauss JG, Olefsky JM. A Gpr120-selective agonist improves insulin resistance and chronic inflammation in obese mice. Nat Med 2014; 20(8):942-947.
- 57. Snodgrass RG, Huang S, Choi IW, Rutledge JC, Hwang DH. Inflammasome-mediated secretion of IL-1beta in human monocytes through TLR2 activation; modulation by dietary fatty acids. J Immunol 2013; 191(8):4337-4347. PMCID: PMC3825708
- 58. Forbes SC, Little JP, Candow DG. Exercise and nutritional interventions for improving aging muscle health. Endocrine 2012; 42(1):29-38.
- 59. Deldicque L, Cani PD, Philp A, Raymackers JM, Meakin PJ, Ashford ML, Delzenne NM, Francaux M, Baar K. The unfolded protein response is activated in skeletal muscle by high-fat feeding: potential role in the downregulation of protein synthesis. Am J Physiol Endocrinol Metab 2010; 299(5):E695-E705.
- 60. Raphael W, Sordillo LM. Dietary polyunsaturated fatty acids and inflammation: the role of phospholipid biosynthesis. Int J Mol Sci 2013; 14(10):21167-21188. PMCID: PMC3821664
- 61. Smith GI, Atherton P, Reeds DN, Mohammed BS, Rankin D, Rennie MJ, Mittendorfer B. Dietary omega-3 fatty acid supplementation increases the rate of muscle protein synthesis in older adults: a randomized controlled trial. Am J Clin Nutr 2011; 93(2):402-412. PMCID: PMC3021432
- 62. Li K, Huang T, Zheng J, Wu K, Li D. Effect of marine-derived n-3 polyunsaturated fatty acids on C-reactive protein, interleukin 6 and tumor necrosis factor alpha: a meta-analysis. PLoS ONE 2014; 9(2):e88103. PMCID: PMC3914936
- 63. Koh EJ, Yoon SJ, Lee SM. Losartan protects liver against ischaemia/reperfusion injury through PPAR-gamma activation and receptor for advanced glycation end-products down-regulation. Br J Pharmacol 2013; 169(6):1404-1416. PMCID: PMC3831716
- 64. An J, Nakajima T, Kuba K, Kimura A. Losartan inhibits LPS-induced inflammatory signaling through a PPARgamma-dependent mechanism in human THP-1 macrophages. Hypertens Res 2010; 33(8):831-835.
- 65. Trevelyan J, Brull DJ, Needham EW, Montgomery HE, Morris A, Mattu RK. Effect of enalapril and losartan on cytokines in patients with stable angina pectoris awaiting coronary artery bypass grafting and their interaction with polymorphisms in the interleukin-6 gene. Am J Cardiol 2004; 94(5):564-569.
- 66. Lin CH, Yang H, Xue QL, Chuang YF, Roy CN, Abadir P, Walston JD. Losartan improves measures of activity, inflammation, and oxidative stress in older mice. Exp Gerontol 2014.
- 67. Kim JE, Choi HC. Losartan Inhibits Vascular Smooth Muscle Cell Proliferation through Activation of AMP-Activated Protein Kinase. Korean J Physiol Pharmacol 2010; 14(5):299-304. PMCID: PMC2997415
- 68. Grossin N, Boulanger E, Wautier MP, Wautier JL. The different isoforms of the receptor for advanced glycation end products are modulated by pharmacological agents. Clin Hemorheol Microcirc 2010; 45(2-4):143-153.
- 69. Burks TN, Andres-Mateos E, Marx R, Mejias R, Van EC, Simmers JL, Walston JD, Ward CW, Cohn RD. Losartan restores skeletal muscle remodeling and protects against disuse atrophy in sarcopenia. Sci Transl Med 2011; 3(82):82ra37. PMCID: PMC3140459

- 70. de GM, Catt KJ, Inagami T, Wright JW, Unger T. International union of pharmacology. XXIII. The angiotensin II receptors. Pharmacol Rev 2000; 52(3):415-472.
- 71. Siddiqui RA, Shaikh SR, Sech LA, Yount HR, Stillwell W, Zaloga GP. Omega 3-fatty acids: health benefits and cellular mechanisms of action. Mini Rev Med Chem 2004; 4(8):859-871.
- 72. Calder PC. Mechanisms of action of (n-3) fatty acids. J Nutr 2012; 142(3):592S-599S.
- 73. Cerreta F, Eichler HG, Rasi G. Drug policy for an aging population--the European Medicines Agency's geriatric medicines strategy. N Engl J Med 2012; 367(21):1972-1974.
- 74. Jeffery CA, Shum DW, Hubbard RE. Emerging drug therapies for frailty. Maturitas 2013; 74(1):21-25.
- 75. Moertl D, Hammer A, Steiner S, Hutuleac R, Vonbank K, Berger R. Dose-dependent effects of omega-3-polyunsaturated fatty acids on systolic left ventricular function, endothelial function, and markers of inflammation in chronic heart failure of nonischemic origin: a double-blind, placebo-controlled, 3-arm study. Am Heart J 2011; 161(5):915-919.
- 76. Nodari S, Triggiani M, Campia U, Manerba A, Milesi G, Cesana BM, Gheorghiade M, Dei CL. Effects of n-3 polyunsaturated fatty acids on left ventricular function and functional capacity in patients with dilated cardiomyopathy. J Am Coll Cardiol 2011; 57(7):870-879.
- 77. Pavlatou MG, Mastorakos G, Margeli A, Kouskouni E, Tentolouris N, Katsilambros N, Chrousos GP, Papassotiriou I. Angiotensin blockade in diabetic patients decreases insulin resistance-associated low-grade inflammation. Eur J Clin Invest 2011; 41(6):652-658.
- 78. Link A, Lenz M, Legner D, Bohm M, Nickenig G. Telmisartan inhibits beta2-integrin MAC-1 expression in human T-lymphocytes. J Hypertens 2006; 24(9):1891-1898.
- 79. Nakamura T, Sato E, Fujiwara N, Kawagoe Y, Yamada S, Ueda Y, Koide H. Changes in urinary albumin excretion, inflammatory and oxidative stress markers in ADPKD patients with hypertension. Am J Med Sci 2012; 343(1):46-51.
- 80. Dahlof B, Devereux RB, Kjeldsen SE, Julius S, Beevers G, de FU, Fyhrquist F, Ibsen H, Kristiansson K, Lederballe-Pedersen O, Lindholm LH, Nieminen MS, Omvik P, Oparil S, Wedel H. Cardiovascular morbidity and mortality in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE): a randomised trial against atenolol. Lancet 2002; 359(9311):995-1003.
- 81. CONSENSUS Trial Study Group. Effects of enalapril on mortality in severe congestive heart failure. Results of the Cooperative North Scandinavian Enalapril Survival Study (CONSENSUS). N Engl J Med 1987; 316:1429-1435.
- 82. Thomas GN, Chan P, Tomlinson B. The role of angiotensin II type 1 receptor antagonists in elderly patients with hypertension. Drugs Aging 2006; 23(2):131-155.
- 83. Pitt B, Segal R, Martinez FA, Meurers G, Cowley AJ, Thomas I, Deedwania PC, Ney DE, Snavely DB, Chang PI. Randomised trial of losartan versus captopril in patients over 65 with heart failure (Evaluation of Losartan in the Elderly Study, ELITE). Lancet 1997; 349:747-752.
- 84. Pitt B, Poole-Wilson PA, Segal R, Martinez FA, Dickstein K, Camm AJ, Konstam MA, Riegger G, Klinger GH, Neaton J, Sharma D, Thiyagarajan B. Effect of losartan compared with captopril on mortality in patients with symptomatic heart failure: randomised trial--the Losartan Heart Failure Survival Study ELITE II. Lancet 2000; 355(9215):1582-1587.

- 85. Marketou ME, Zacharis EA, Koukouraki S, Stathaki MI, Arfanakis DA, Kochiadakis GE, Chlouverakis G, Karkavitsas NS, Vardas PE. Effect of angiotensin-converting enzyme inhibitors on systemic inflammation and myocardial sympathetic innervation in normotensive patients with type 2 diabetes mellitus. J Hum Hypertens 2008; 22(3):191-196.
- 86. Madej A, Buldak L, Basiak M, Szkrobka W, Dulawa A, Okopien B. The effects of 1 month antihypertensive treatment with perindopril, bisoprolol or both on the ex vivo ability of monocytes to secrete inflammatory cytokines. Int J Clin Pharmacol Ther 2009; 47(11):686-694.
- 87. Sumukadas D, Witham MD, Struthers AD, McMurdo ME. Effect of perindopril on physical function in elderly people with functional impairment: a randomized controlled trial. CMAJ 2007; 177(8):867-874.
- 88. Koz C, Baysan O, Yokusoglu M, Uzun M, Yildirim M, Hasimi A, Oz BS, Erinc K, Karaeren H, Celebi H, Isik E. The effects of perindopril on aortic elasticity and inflammatory markers in hypertensive patients. Med Sci Monit 2009; 15(7):I41-I45.
- 89. Randomised trial of a perindopril-based blood-pressure-lowering regimen among 6,105 individuals with previous stroke or transient ischaemic attack. Lancet 2001; 358(9287):1033-1041.
- 90. Makani H, Bangalore S, Desouza KA, Shah A, Messerli FH. Efficacy and safety of dual blockade of the renin-angiotensin system: meta-analysis of randomised trials. BMJ 2013; 346:f360. PMCID: PMC3556933
- 91. Derosa G, Maffioli P, Salvadeo SA, Ferrari I, Gravina A, Mereu R, Palumbo I, D'Angelo A, Cicero AF. Candesartan effect on inflammation in hypertension. Hypertens Res 2010; 33(3):209-213.
- 92. Sola S, Mir MQ, Cheema FA, Khan-Merchant N, Menon RG, Parthasarathy S, Khan BV. Irbesartan and lipoic acid improve endothelial function and reduce markers of inflammation in the metabolic syndrome: results of the Irbesartan and Lipoic Acid in Endothelial Dysfunction (ISLAND) study. Circulation 2005; 111(3):343-348.
- 93. Persson F, Rossing P, Hovind P, Stehouwer CD, Schalkwijk C, Tarnow L, Parving HH. Irbesartan treatment reduces biomarkers of inflammatory activity in patients with type 2 diabetes and microalbuminuria: an IRMA 2 substudy. Diabetes 2006; 55(12):3550-3555.
- 94. Ceriello A, Assaloni R, Da RR, Maier A, Piconi L, Quagliaro L, Esposito K, Giugliano D. Effect of atorvastatin and irbesartan, alone and in combination, on postprandial endothelial dysfunction, oxidative stress, and inflammation in type 2 diabetic patients. Circulation 2005; 111(19):2518-2524.
- 95. Schieffer B, Bunte C, Witte J, Hoeper K, Boger RH, Schwedhelm E, Drexler H. Comparative effects of AT1-antagonism and angiotensin-converting enzyme inhibition on markers of inflammation and platelet aggregation in patients with coronary artery disease. J Am Coll Cardiol 2004; 44(2):362-368.
- 96. Nakayama S, Watada H, Mita T, Ikeda F, Shimizu T, Uchino H, Fujitani Y, Hirose T, Kawamori R. Comparison of effects of olmesartan and telmisartan on blood pressure and metabolic parameters in Japanese early-stage type-2 diabetics with hypertension. Hypertens Res 2008; 31(1):7-13.
- 97. Takagi H, Mizuno Y, Yamamoto H, Goto SN, Umemoto T. Effects of telmisartan therapy on interleukin-6 and tumor necrosis factor-alpha levels: a meta-analysis of randomized controlled trials. Hypertens Res 2013; 36(4):368-373.

- 98. Hong SJ, Shim WJ, Choi JI, Joo HJ, Shin SY, Park SM, Lim SY, Lim DS. Comparison of effects of telmisartan and valsartan on late lumen loss and inflammatory markers after sirolimus-eluting stent implantation in hypertensive patients. Am J Cardiol 2007; 100(11):1625-1629.
- 99. Janic M, Lunder M, Prezelj M, Sabovic M. A combination of low-dose fluvastatin and valsartan decreases inflammation and oxidative stress in apparently healthy middle-aged males. J Cardiopulm Rehabil Prev 2014; 34(3):208-212.
- 100. Kintscher U, Marx N, Martus P, Stoppelhaar M, Schimkus J, Schneider A, Walcher D, Kummel A, Winkler R, Kappert K, Dorffel Y, Scholze J, Unger T. Effect of high-dose valsartan on inflammatory and lipid parameters in patients with Type 2 diabetes and hypertension. Diabetes Res Clin Pract 2010; 89(3):209-215.
- 101. Manabe S, Okura T, Watanabe S, Fukuoka T, Higaki J. Effects of angiotensin II receptor blockade with valsartan on pro-inflammatory cytokines in patients with essential hypertension. J Cardiovasc Pharmacol 2005; 46(6):735-739.
- 102. Touyz RM, Savoia C, He Y, Endemann D, Pu Q, Ko EA, Deciuceis C, Montezano A, Schiffrin EL. Increased inflammatory biomarkers in hypertensive type 2 diabetic patients: improvement after angiotensin II type 1 receptor blockade. J Am Soc Hypertens 2007; 1(3):189-199.
- 103. Zankl AR, Ivandic B, Andrassy M, Volz HC, Krumsdorf U, Blessing E, Katus HA, Tiefenbacher CP. Telmisartan improves absolute walking distance and endothelial function in patients with peripheral artery disease. Clin Res Cardiol 2010; 99(12):787-794.
- 104. Caldeira D, David C, Sampaio C. Tolerability of angiotensin-receptor blockers in patients with intolerance to angiotensin-converting enzyme inhibitors: a systematic review and meta-analysis. Am J Cardiovasc Drugs 2012; 12(4):263-277.
- 105. Zhang Y, Han P, Wu N, He B, Lu Y, Li S, Liu Y, Zhao S, Liu L, Li Y. Amelioration of lipid abnormalities by alpha-lipoic acid through antioxidative and anti-inflammatory effects. Obesity (Silver Spring) 2011; 19(8):1647-1653.
- 106. Mollo R, Zaccardi F, Scalone G, Scavone G, Rizzo P, Navarese EP, Manto A, Pitocco D, Lanza GA, Ghirlanda G, Crea F. Effect of alpha-lipoic acid on platelet reactivity in type 1 diabetic patients. Diabetes Care 2012; 35(2):196-197. PMCID: PMC3263886
- 107. Hutchins-Wiese HL, Kleppinger A, Annis K, Liva E, Lammi-Keefe CJ, Durham HA, Kenny AM. The impact of supplemental n-3 long chain polyunsaturated fatty acids and dietary antioxidants on physical performance in postmenopausal women. J Nutr Health Aging 2013; 17(1):76-80.
- 108. Rodacki CL, Rodacki AL, Pereira G, Naliwaiko K, Coelho I, Pequito D, Fernandes LC. Fish-oil supplementation enhances the effects of strength training in elderly women. Am J Clin Nutr 2012; 95(2):428-436.
- 109. Schwingshackl L, Hoffmann G. Mediterranean dietary pattern, inflammation and endothelial function: A systematic review and meta-analysis of intervention trials. Nutr Metab Cardiovasc Dis 2014.
- 110. Casas R, Sacanella E, Urpi-Sarda M, Chiva-Blanch G, Ros E, Martinez-Gonzalez MA, Covas MI, Salas-Salvado J, Fiol M, Aros F, Estruch R. The effects of the mediterranean diet on biomarkers of vascular wall inflammation and plaque vulnerability in subjects with high risk for cardiovascular disease. A randomized trial. PLoS ONE 2014; 9(6):e100084. PMCID: PMC4055759

- 111. Urpi-Sarda M, Casas R, Chiva-Blanch G, Romero-Mamani ES, Valderas-Martinez P, Arranz S, Andres-Lacueva C, Llorach R, Medina-Remon A, Lamuela-Raventos RM, Estruch R. Virgin olive oil and nuts as key foods of the Mediterranean diet effects on inflammatory biomakers related to atherosclerosis. PHARMACOL RES 2012; 65(6):577-583.
- 112. Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med 2006; 145(1):1-11.
- 113. Esposito K, Marfella R, Ciotola M, Di PC, Giugliano F, Giugliano G, D'Armiento M, D'Andrea F, Giugliano D. Effect of a mediterranean-style diet on endothelial dysfunction and markers of vascular inflammation in the metabolic syndrome: a randomized trial. JAMA 2004; 292(12):1440-1446.
- 114. Beauchamp GK, Keast RS, Morel D, Lin J, Pika J, Han Q, Lee CH, Smith AB, Breslin PA. Phytochemistry: ibuprofen-like activity in extra-virgin olive oil. Nature 2005; 437(7055):45-46.
- 115. Zbeida M, Goldsmith R, Shimony T, Vardi H, Naggan L, Shahar DR. Mediterranean diet and functional indicators among older adults in non-Mediterranean and Mediterranean countries. J Nutr Health Aging 2014; 18(4):411-418.
- 116. Talegawkar SA, Bandinelli S, Bandeen-Roche K, Chen P, Milaneschi Y, Tanaka T, Semba RD, Guralnik JM, Ferrucci L. A higher adherence to a Mediterranean-style diet is inversely associated with the development of frailty in community-dwelling elderly men and women. J Nutr 2012; 142(12):2161-2166. PMCID: PMC3497964
- 117. Bollwein J, Diekmann R, Kaiser MJ, Bauer JM, Uter W, Sieber CC, Volkert D. Dietary quality is related to frailty in community-dwelling older adults. J Gerontol A Biol Sci Med Sci 2013; 68(4):483-489.
- 118. Shahar DR, Houston DK, Hue TF, Lee JS, Sahyoun NR, Tylavsky FA, Geva D, Vardi H, Harris TB. Adherence to mediterranean diet and decline in walking speed over 8 years in community-dwelling older adults. J Am Geriatr Soc 2012; 60(10):1881-1888. PMCID: PMC3470771
- 119. Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med 2013; 368(14):1279-1290.
- 120. Bongartz T, Sutton AJ, Sweeting MJ, Buchan I, Matteson EL, Montori V. Anti-TNF antibody therapy in rheumatoid arthritis and the risk of serious infections and malignancies: systematic review and metaanalysis of rare harmful effects in randomized controlled trials. JAMA 2006; 295(19):2275-2285.
- 121. Voorhees PM, Manges RF, Sonneveld P, Jagannath S, Somlo G, Krishnan A, Lentzsch S, Frank RC, Zweegman S, Wijermans PW, Orlowski RZ, Kranenburg B, Hall B, Casneuf T, Qin X, van d, V, Xie H, Thomas SK. A phase 2 multicentre study of siltuximab, an anti-interleukin-6 monoclonal antibody, in patients with relapsed or refractory multiple myeloma. Br J Haematol 2013; 161(3):357-366.
- 122. Howard C, Noe A, Skerjanec A, Holzhauer B, Wernsing M, Ligueros-Saylan M, Thuren T. Safety and tolerability of canakinumab, an IL-1beta inhibitor, in type 2 diabetes mellitus patients: a pooled analysis of three randomised double-blind studies. Cardiovasc Diabetol 2014; 13:94. PMCID: PMC4033489

- 123. Singh S, Loke YK, Furberg CD. Long-term use of thiazolidinediones and the associated risk of pneumonia or lower respiratory tract infection: systematic review and meta-analysis. Thorax 2011; 66(5):383-388.
- 124. Norata GD, Tibolla G, Catapano AL. Statins and skeletal muscles toxicity: From clinical trials to everyday practice. PHARMACOL RES 2014.
- 125. Avina-Zubieta JA, Johnson ES, Suarez-Almazor ME, Russell AS. Incidence of myopathy in patients treated with antimalarials. A report of three cases and a review of the literature. Br J Rheumatol 1995; 34(2):166-170.
- 126. Oyama F, Murakami N, Ihara Y. Chloroquine myopathy suggests that tau is degraded in lysosomes: implication for the formation of paired helical filaments in Alzheimer's disease. Neurosci Res 1998; 31(1):1-8.
- 127. Parker BA, Capizzi JA, Grimaldi AS, Clarkson PM, Cole SM, Keadle J, Chipkin S, Pescatello LS, Simpson K, White CM, Thompson PD. Effect of statins on skeletal muscle function. Circulation 2013; 127(1):96-103.
- 128. Yuhara H, Corley DA, Nakahara F, Nakajima T, Koike J, Igarashi M, Suauki T, Mine T. Aspirin and non-aspirin NSAIDs increase risk of colonic diverticular bleeding: a systematic review and meta-analysis. J Gastroenterol 2014; 49(6):992-1000.
- 129. Jarupongprapa S, Ussavasodhi P, Katchamart W. Comparison of gastrointestinal adverse effects between cyclooxygenase-2 inhibitors and non-selective, non-steroidal anti-inflammatory drugs plus proton pump inhibitors: a systematic review and meta-analysis. J Gastroenterol 2013; 48(7):830-838.
- 130. Wang X, Tian HJ, Yang HK, Wanyan P, Peng YJ. Meta-analysis: cyclooxygenase-2 inhibitors are no better than nonselective nonsteroidal anti-inflammatory drugs with proton pump inhibitors in regard to gastrointestinal adverse events in osteoarthritis and rheumatoid arthritis. Eur J Gastroenterol Hepatol 2011; 23(10):876-880.
- 131. Narum S, Westergren T, Klemp M. Corticosteroids and risk of gastrointestinal bleeding: a systematic review and meta-analysis. BMJ Open 2014; 4(5):e004587. PMCID: PMC4025450
- 132. Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet 2009; 373(9678):1849-1860. PMCID: PMC2715005
- 133. Hennekens CH, Borzak S. Cyclooxygenase-2 inhibitors and most traditional nonsteroidal antiinflammatory drugs cause similar moderately increased risks of cardiovascular disease. J Cardiovasc Pharmacol Ther 2008; 13(1):41-50.
- 134. Ching JK, Ju JS, Pittman SK, Margeta M, Weihl CC. Increased autophagy accelerates colchicine-induced muscle toxicity. Autophagy 2013; 9(12):2115-2125.
- 135. Kuncl RW, Duncan G, Watson D, Alderson K, Rogawski MA, Peper M. Colchicine myopathy and neuropathy. N Engl J Med 1987; 316(25):1562-1568.
- 136. Haffner S, Temprosa M, Crandall J, Fowler S, Goldberg R, Horton E, Marcovina S, Mather K, Orchard T, Ratner R, Barrett-Connor E. Intensive lifestyle intervention or metformin on inflammation and

- coagulation in participants with impaired glucose tolerance. Diabetes 2005; 54(5):1566-1572. PMCID: PMC1314967
- 137. Erem C, Ozbas HM, Nuhoglu I, Deger O, Civan N, Ersoz HO. Comparison of effects of gliclazide, metformin and pioglitazone monotherapies on glycemic control and cardiovascular risk factors in patients with newly diagnosed uncontrolled type 2 diabetes mellitus. Exp Clin Endocrinol Diabetes 2014; 122(5):295-302.
- 138. Kadoglou NP, Kapelouzou A, Tsanikidis H, Vitta I, Liapis CD, Sailer N. Effects of rosiglitazone/metformin fixed-dose combination therapy and metformin monotherapy on serum vaspin, adiponectin and IL-6 levels in drug-naive patients with type 2 diabetes. Exp Clin Endocrinol Diabetes 2011; 119(2):63-68.
- 139. Kim HJ, Kang ES, Kim DJ, Kim SH, Ahn CW, Cha BS, Nam M, Chung CH, Lee KW, Nam CM, Lee HC. Effects of rosiglitazone and metformin on inflammatory markers and adipokines: decrease in interleukin-18 is an independent factor for the improvement of homeostasis model assessment-beta in type 2 diabetes mellitus. Clin Endocrinol (Oxf) 2007; 66(2):282-289.
- 140. Gomez-Diaz RA, Talavera JO, Pool EC, Ortiz-Navarrete FV, Solorzano-Santos F, Mondragon-Gonzalez R, Valladares-Salgado A, Cruz M, Aguilar-Salinas CA, Wacher NH. Metformin decreases plasma resistin concentrations in pediatric patients with impaired glucose tolerance: a placebo-controlled randomized clinical trial. Metabolism 2012; 61(9):1247-1255.
- 141. Deans KA, Sattar N. "Anti-inflammatory" drugs and their effects on type 2 diabetes. Diabetes Technol Ther 2006; 8(1):18-27.
- 142. Pradhan AD, Everett BM, Cook NR, Rifai N, Ridker PM. Effects of initiating insulin and metformin on glycemic control and inflammatory biomarkers among patients with type 2 diabetes: the LANCET randomized trial. JAMA 2009; 302(11):1186-1194.
- 143. Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD. Effect of Structured Physical Activity on Prevention of Major Mobility Disability in Older Adults: The LIFE Study Randomized Clinical Trial. JAMA 2014; 311(23):2387-2396. PMCID: 24866862
- 144. LIFE investigators, Pahor M, Blair SN, Espeland M, Fielding RA, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a Physical Activity Intervention on Measures of Physical Performance: Results of the Lifestyle Interventions and Independence for Elders Pilot (LIFE-P) Study. J Gerontol A Biol Sci Med Sci 2006; 61(11):1157-1165. PMCID: PMID:17167156
- 145. Messier SP, Miller GD, Morgan TP, Rejeski WJ, Sevick MA, Loeser RF, Ettinger WH, Pahor M, Williamson JD. Exercise and dietary weight loss in overweight and obese older adults with knee osteoarthritis: the Arthritis, Diet and Activity Promotion Trial (ADAPT). Arthritis and Rheumatism 2004; 50:1501-1510.
- 146. Villareal DT, Chode S, Parimi N, Sinacore DR, Hilton T, Armamento-Villareal R, Napoli N, Qualls C, Shah K. Weight loss, exercise, or both and physical function in obese older adults. N Engl J Med 2011; 364(13):1218-1229. PMCID: PMC3114602

- 147. Anton SD, Manini TM, Milson V, Dubyak P, Cesari M, Cheng J, Daniels MJ, Marsiske M, Pahor M, Leeuwenburgh CL, Perri MG. Effects of a weight loss plus exercise program on physical functioning in overweight, older women: a randomized controlled trial. Clinical Interventions in Aging 2011; 6:141-149.
- 148. Villani AM, Crotty M, Cleland LG, James MJ, Fraser RJ, Cobiac L, Miller MD. Fish oil administration in older adults: is there potential for adverse events? A systematic review of the literature. BMC Geriatr 2013; 13(1):41. PMCID: PMC3664575
- 149. Villani AM, Crotty M, Cleland LG, James MJ, Fraser RJ, Cobiac L, Miller MD. Fish oil administration in older adults with cardiovascular disease or cardiovascular risk factors: is there potential for adverse events? A systematic review of the literature. Int J Cardiol 2013; 168(4):4371-4375.
- 150. Sakkinen PA, Macy EM, Callas PW, Cornell ES, Hayes TE, Kuller LH, Tracy RP. Analytical and biologic variability in measures of hemostasis, fibrinolysis, and inflammation: assessment and implications for epidemiology. Am J Epidemiol 1999; 149(3):261-267.
- 151. Knudsen LS, Christensen IJ, Lottenburger T, Svendsen MN, Nielsen HJ, Nielsen L, Horslev-Petersen K, Jensen JE, Kollerup G, Johansen JS. Pre-analytical and biological variability in circulating interleukin 6 in healthy subjects and patients with rheumatoid arthritis. Biomarkers 2008; 13(1):59-78.
- 152. King MA, Pryce RL. Evidence for compliance with long-term medication: a systematic review of randomised controlled trials. Int J Clin Pharm 2014; 36(1):128-135.
- 153. Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav 2008; 12(1):86-94.
- 154. Cesari M, Kritchevsky SB, Penninx BWJH, Nicklas BJ, Simonsick EM, Newman AB, Tylavsky F, Brach JS, Satterfield S, Bauer DC, Visser M, Rubin S, Harris TB, Pahor M. Prognostic value of usual gait speed in well-functioning older people-results from the health, aging and body composition study. J Am Geriatr Soc 2005; 53:1675-1680.
- 155. Cesari M, Kritchevsky SB, Newman AB, Simonsick EM, Harris TB, Penninx BW, Brach JS, Tylavsky FA, Satterfield S, Bauer DC, Rubin SM, Visser M, Pahor M. Added value of physical performance measures in predicting adverse health-related events: results from the Health, Aging And Body Composition Study. J Am Geriatr Soc 2009; 57(2):251-259.
- 156. Picotte M, Campbell CG, Thorland WG. Day-to-day variation in plasma interleukin-6 concentrations in older adults. Cytokine 2009; 47(3):162-165.
- 157. Marsh AP, Lovato LC, Glynn NW, Kennedy K, Castro C, Domanchuk K, McDavitt E, Rodate R, Marsiske M, McGloin J, Groessl EJ, Pahor M, Guralnik JM. Lifestyle Interventions and Independence for Elders Study: Recruitment and Baseline Characteristics. J Gerontol A Biol Sci Med Sci 2013; 68(12):1549-1558. PMCID: PMC3814232
- 158. Katula JA, Kritchevsky SB, Guralnik JM, Glynn NW, Pruitt L, Wallace K, Walkup MP, Hsu FC, Studenski SA, Gill TM, Groessl EJ, Wallace JM, Pahor M. Lifestyle interventions and independence for elders pilot study: recruitment and baseline characteristics. J Am Geriatr Soc 2007; 55(5):674-683. PMCID: PMID:17493186
- 159. Snyder PJ, Ellenberg SS, Cunningham GR, Matsumoto AM, Bhasin S, Barrett-Connor E, Gill TM, Farrar JT, Cella D, Rosen RC, Resnick SM, Swerdloff RS, Cauley JA, Cifelli D, Fluharty L, Pahor M, Ensrud KE, Lewis CE, Molitch ME, Crandall JP, Wang C, Budoff MJ, Wenger NK, Mohler ER, III, Bild DE, Cook NL, Keaveny TM, Kopperdahl DL, Lee D, Schwartz AV, Storer TW, Ershler WB, Roy CN,

- Raffel LJ, Romashkan S, Hadley E. The Testosterone Trials: Seven coordinated trials of testosterone treatment in elderly men. Clin Trials 2014; 11(3):362-375.
- 160. Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab 2011; 96(1):53-58. PMCID: PMC3046611
- 161. Parving HH, Brenner BM, McMurray JJ, de ZD, Haffner SM, Solomon SD, Chaturvedi N, Persson F, Desai AS, Nicolaides M, Richard A, Xiang Z, Brunel P, Pfeffer MA. Cardiorenal end points in a trial of aliskiren for type 2 diabetes. N Engl J Med 2012; 367(23):2204-2213.
- 162. Fielding RA, Rejeski WJ, Blair SN, Church T, Espeland MA, Guralnik JM, Gill TM, Hsu FC, Katula JA, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds DE, Romashkan S, Hadley E, Pahor M. The Lifestyle Interventions and Independence for Elders (LIFE) Study: Design and Methods. J Gerontol A Biol Sci Med Sci 2011; 66(11):1226-1237. PMCID: PMC3193523
- 163. Brault MW. Americans With Disabilities: 2010 Household Economic Studies. Current Population Reports. U.S. CENSUS BUREAU U.S. Department of Commerce Economics and Statistics Administration; 2012 p. 70-131.
- 164. Rolland YM, Cesari M, Miller ME, Penninx BWJH, Atkinson H, Pahor M. Reliability of the 400-meter usual pace walk test as an assessment of mobility limitation in older adults. J Am Geriatr Soc 2004; 52:972-976.
- 165. Lonergan ET, Krevans JR. A national agenda for research on aging. N Engl J Med 1991; 324(25):1825-1828
- Guralnik JM, LaCroix AZ, Abbott RD, Berkman LF, Satterfield S, Evans DA, Wallace RB. Maintaining mobility in late life. I. Demographic characteristics and chronic conditions. Am J Epidemiol 1993; 137:845-857.
- 167. Espeland MA, Gill TM, Guralnik JM, Miller ME, Fielding RA, Newman AB, Pahor M. Designing Clinical Trials of Intervention for Mobility Disability: results from the Lifestyle Interventions and Independence for Elders (LIFE) Pilot trial. J Gerontol A Biol Sci Med Sci 2007; 62(11):1237-1243. PMCID: PMC2376827
- 168. Hoxie RE, Rubenstein LZ. Are older pedestrians allowed enough time to cross intersections safely? J Am Geriatr Soc 1994; 42(3):241-244.
- 169. Fiatarone MA. Elderly patients and frailty. Resistance training for health and rehabilitation. Champaign IL: Human Kinetics; 2001 p. 181-213.
- 170. Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci 2001; 56(3):M146-M156.
- 171. Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci 2001; 56(3):M146-M156.

- 172. Rantanen T, Harris T, Leveille SG, Visser M, Foley D, Masaki K, Guralnik JM. Muscle strength and body mass index as long-term predictors of mortality in initially healthy men. J Gerontol A Biol Sci Med Sci 2000; 55(3):M168-M173.
- 173. Rantanen T, Guralnik JM, Foley D, Masaki K, Leveille S, Curb JD, White L. Midlife hand grip strength as a predictor of old age disability. JAMA 1999; 281(6):558-560.
- 174. Visser M, Pahor M, Taaffe D, Goodpaster BH, Simonsick E, Newman AB, Nevitt MC, Harris TB. Relationship of interleukin-6 and tumor necrosis factor-á with muscle mass and muscle strength in elderly men and women: the Health ABC Study. J Gerontol A Biol Sci Med Sci 2002; 57:M326-M332.
- 175. Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. Appl Psychol Measurement 1977; 1(3):385-401.
- 176. Manini TM, Visser M, Won-Park S, Patel KV, Strotmeyer ES, Chen H, Goodpaster B, de RN, Newman AB, Simonsick EM, Kritchevsky SB, Ryder K, Schwartz AV, Harris TB. Knee extension strength cutpoints for maintaining mobility. J Am Geriatr Soc 2007; 55(3):451-457.
- 177. Molczyk L, Thigpen LK, Eickhoff J, Goldgar D, Gallagher JC. Reliability of Testing the Knee Extensors and Flexors in Healthy Adult Women Using a Cybex II Isokinetic Dynamometer. J Orthop Sports Phys Ther 1991; 14(1):37-41.
- 178. Friedlander AL, Block JE, Byl NN, Stubbs HA, Sadowsky HS, Genant HK. Isokinetic limb and trunk muscle performance testing: short-term reliability. J Orthop Sports Phys Ther 1991; 14(5):220-224.
- 179. Ebid AA, Ahmed MT, Mahmoud EM, Mohamed MS. Effect of whole body vibration on leg muscle strength after healed burns: a randomized controlled trial. Burns 2012; 38(7):1019-1026.
- 180. Ly LP, Jimenez M, Zhuang TN, Celermajer DS, Conway AJ, Handelsman DJ. A double-blind, placebo-controlled, randomized clinical trial of transdermal dihydrotestosterone gel on muscular strength, mobility, and quality of life in older men with partial androgen deficiency. J Clin Endocrinol Metab 2001; 86(9):4078-4088.
- McHorney CA, Ware JE, Jr., Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care 1994; 32(1):40-66.
- 182. McHorney CA, Ware JE, Jr., Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care 1993; 31(3):247-263.
- 183. Snow KK, Snow KK, Kosinski M, Gandek B. SF-36 Health survey manual and interpretation guide. Boston: The Health Institute, New England Medical Center; 1993.
- 184. Ware JE, Jr., Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care 1992; 30(6):473-483.
- 185. Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res 1975; 12(3):189-198.
- 186. Taylor HL, Jacobs DR, Jr., Schucker B, Knudsen J, Leon AS, Debacker G. A questionnaire for the assessment of leisure time physical activities. J Chronic Dis 1978; 31(12):741-755.

- 187. Rubinstein LV, Korn EL, Freidlin B, Hunsberger S, Ivy SP, Smith MA. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol 2005; 23(28):7199-7206.
- 188. Hunsberger S, Zhao Y, Simon R. A comparison of phase II study strategies. Clin Cancer Res 2009; 15(19):5950-5955. PMCID: PMC2757284
- 189. FDA Code of Federal Regulations. TITLE 21--FOOD AND DRUGSCHAPTER I--FOOD AND DRUG ADMINISTRATION DEPARTMENT OF HEALTH AND HUMAN SERVICES SUBCHAPTER D--DRUGS FOR HUMAN USE PART 312 -- INVESTIGATIONAL NEW DRUG APPLICATION Subpart B-Investigational New Drug Application (IND). Title 21, Volume 5 ed. 2014.
- 190. The FDA's Drug Review Process: Ensuring Drugs Are Safe and Effective Accessed on 9/19/1014 http://www.fda.gov/drugs/resourcesforyou/consumers/ucm143534.htm. 2014.
- 191. Fay MP. Confidence intervals that match Fisher's exact or Blaker's exact tests. Biostatistics 2010; 11(2):373-374. PMCID: PMC2852239
- 192. Kwon S, Perera S, Pahor M, Katula JA, King AC, Groessl EJ, Studenski S. What is a meaningful change in physical performance? findings from a clinical trial in older adults (the LIFE-P study). J Nutr Health Aging 2009; 13(6):538-544. PMCID: PMC3100159
- 193. Proschan MA, Lan KKG, Wittes JT. Statistical Monitoring of Clincial Trials, A Unified Approach. New York, NY: Springer Science; 2006.
- 194. SHEP Cooperative Research Group. Prevention of stroke by antihypertensive drug treatment in older persons with isolated systolic hypertension. Final results of the Systolic Hypertension in the Elderly Program (SHEP). JAMA 1991; 265:3255-3264.
- 195. Fried LP, Borhani NO, Enright P, Furberg CD, Gardin JM, Kronmal RA, Kuller LH, Manolio TA, Mittelmark MB, Newman A, et al. The Cardiovascular Health Study: design and rationale. Ann Epidemiol 1991; 1(3):263-276.
- 196. Simonsick EM, Montgomery PS, Newman AB, Bauer DC, Harris T. Measuring fitness in healthy older adults: the Health ABC Long Distance Corridor Walk. J Am Geriatr Soc 2001; 49(11):1544-1548.
- 197. The Women's Health and Aging Study. Health and social characteristics of older women with disability. Bethesda: National Institute on Aging. NIH publication No. 95-4009; 1995.
- 198. Glynn NW, Santanasto AJ, Simonsick EM, Boudreau RM, Beach SR, Schulz R, Newman AB. The Pittsburgh Fatigability scale for older adults: development and validation. J Am Geriatr Soc. 2015 Jan;63(1):130-5. doi: 10.1111/jgs.13191. Epub 2014 Dec 31. PubMed PMID: 25556993.